# NCT02247804

Study ID: 192024-091

Title: Efficacy and Safety of Bimatoprost Sustained-Release (SR) in Patients With Open-angle Glaucoma or Ocular Hypertension

Protocol Amendment 2 Date: 16-Mar-2017

# Approval Date: 16-Mar-2017

# ALLERGAN – CONFIDENTIAL

The following contains confidential, proprietary information which is the property of Allergan

# The Efficacy and Safety of Bimatoprost SR in Patients With Open-angle Glaucoma or Ocular Hypertension

Protocol Number: 192024-091 Amendment 2

EudraCT Number: 2014-003037-26

Phase: 3

Name of Investigational Product: Bimatoprost SR

Sponsor: Allergan (North America) Allergan Ltd.
2525 Dupont Drive 1st Floor, Marlow

Irvine, California USA International,

92612

1

+1-714-246-4500 Buckinghamshire

+1-800-347-4500 SL7 1YL United Kingdom

Tel: +44 (0) 1628 494444 Fax: +44 (0) 1628 494449

The Parkway, Marlow

Emergency Telephone Numbers: Refer to the Study Contacts Page.



Allergan Signatory:



Refer to the final page of this protocol for electronic signature and date of approval.

The following information can be found on FDA Form 1572 and/or study contacts page: name and contact information of Allergan study personnel and emergency telephone numbers; name, address, and statement of qualifications of each investigator; name of each subinvestigator working under the supervision of the investigator; name and address of the research facilities to be used; name and address of each reviewing institutional review board (IRB); US 21 CFR 312.23 section 6(iii)b.

## INVESTIGATOR SIGNATURE PAGE

| TNT | EST | $C_{-}I$ | \T | $^{\circ}$ | ρ. |
|-------|-------|----------|----|------------|----|
| TIA A | LO II | CI/ | 71 | V. | Ν. |

## I agree to:

- Implement and conduct this study diligently and in strict compliance with the protocol, good clinical practices and all applicable laws and regulations
- Maintain all information supplied by Allergan in confidence, and when this information
  is submitted to an institutional review board (IRB), independent ethics committee (IEC)
  or another group, it will be submitted with a designation that the material is confidential
- Ensure that all persons assisting with the trial are adequately informed about the protocol, the investigational product(s), and their trial-related duties and functions.

I have read this protocol in its entirety and I agree to all aspects.

| Investigator Printed Name | Signature | Date |
|---------------------------|-----------|------|

# **Table of Contents**

| Tab | le of | Contents | 4 |
|---|---|---|---|
| List | t of Ta | ables | 8 |
| List | t of Fi | igures | 9 |
| Pro | tocol | Summary | 10 |
| 1. | Back | ground and Clinical Rationale | 24 |
| | 1.1 | Glaucoma Overview | |
| | 1.2 | Bimatoprost (LUMIGAN®) | |
| | 1.3 | Bimatoprost SR | |
| | | 1.3.1 Nonclinical Studies with Bimatoprost SR | |
| | | 1.3.2 Other Biodegradable Ocular Implants | |
| | | 1.3.3 Clinical Study with Bimatoprost SR | |
| | 1.4 | Study Rationale | |
| 2. | Stud | y Objectives and Clinical Hypotheses | 29 |
| | 2.1 | Study Objectives | 29 |
| | 2.2 | Clinical Hypotheses | 29 |
| 3. | Stud | y Design | 29 |
| 4. | Stud | y Population and Entry Criteria | 31 |
| | 4.1 | Number of Patients | 31 |
| | 4.2 | Study Population Characteristics | 31 |
| | | 4.2.1 Patients With Sickle Cell Trait or Disease | 31 |
| | 4.3 | Inclusion Criteria | |
| | 4.4 | Exclusion Criteria | 33 |
| | 4.5 | Permissible and Prohibited Medications/Treatments | 37 |
| | | 4.5.1 Permissible Medications/Treatments | 37 |
| | | 4.5.2 Prohibited Medications/Treatments | 38 |
| | | 4.5.3 Definition of Females of (Non-)Childbearing Potential and/or Accepta Contraceptive Methods | |
| 5. | Stud | y Treatments | |
| | 5.1 | Study Treatments and Formulations | |
| | 5.2 | Control Treatments | |
| | 5.3 | Methods for Masking | 41 |
| | 5.4 | Treatment Allocation Ratio and Stratification | 43 |

| | 5.5 | Method for Assignment to Treatment Groups/Randomization | 43 |
|---|---|---|---|
| | 5.6 | Treatment Regimen and Dosing | 44 |
| | | 5.6.1 Treatment Regimen/Dosage Adjustments | 44 |
| | 5.7 | Storage of Study Medications/Treatments | 45 |
| | 5.8 | Preparation of Study Medications/Treatments | 46 |
| | 5.9 | Treatment Administration | 46 |
| | | 5.9.1 Patient Preparation | 46 |
| | | 5.9.2 Study Treatment Location | 46 |
| | | 5.9.3 Administration Technique | <b>4</b> 7 |
| | | 5.9.4 Immediate Posttreatment Observation | <b>4</b> 7 |
| | 5.10 | Retreatment | 48 |
| 6. | Resp | onse Measures and Summary of Data Collection Methods | 48 |
| | 6.1 | Efficacy Measures | 48 |
| | | 6.1.1 Primary Efficacy Measure | 48 |
| | 6.2 | Safety Measures | |
| • | 6.4 | Examination Procedures, Tests, Equipment, and Techniques | 52 |
| | | 6.4.1 Medical History, Physical Examination, and Vital Signs | 52 |
| | | 6.4.1.1 Medical History | |
| | | 6.4.1.2 Physical Examination | 53 |
| | | 6.4.1.3 Vital Signs | 53 |
| | | 6.4.2 Pregnancy Testing | 53 |
| | | 6.4.3 Laboratory Procedures | 53 |
| | | 6.4.3.1 Hematology | 54 |
| | | 6.4.3.2 Serum Chemistry | 54 |
| | | 6.4.3.3 Urinalysis | 54 |
| | 6.5 | Other Study Supplies | 54 |
| | 6.6 | Summary of Methods of Data Collection | 55 |
| 7. | Stati | stical Procedures | 55 |
| | 7.1 | Analysis Populations | 56 |
| | 7.2 | Collection and Derivation of Primary and Secondary Efficacy Assessments | |
| | | 7.2.1 Primary Efficacy Variable | |
| | | 7.2.2 Secondary Efficacy Variable | 57 |
| | 7.3 | Hypothesis and Methods of Analysis | |
| | | 7.3.1 Primary Efficacy Analyses | 57 |

| | | 7.3.2 Secondary Efficacy Analyses 58 |
|----|------|--------------------------------------------|
| | | 7.3.4 Safety Analyses |
| | 7.4 | Subgroup Analyses 59 |
| | 7.5 | Interim Analyses |
| | 7.6 | Analyses for US FDA |
| | 7.7 | Sample Size Calculation |
| 8. | Stud | y Visit Schedule and Procedures |
| | 8.1 | Patient Entry Procedures 62 |
| | | 8.1.1 Overview of Entry Procedures 62 |
| | | 8.1.2 Informed Consent and Patient Privacy |
| | 8.2 | Washout Intervals 62 |
| | 8.3 | Procedures for Final Study Entry |



| 8.5 | Instructions for the Patients | . 82 |
|---|---|---|
| 8.6 | Unscheduled Visits | . 83 |
| 8.7 | | |
| 88 | • | |
| 8.9 | | |
| 8.10 | | |
| | 9.1.2 Serious Adverse Event | |
| | 9.1.3 Severity | |
| | 9.1.4 Relationship to Study Drug or Study Procedure | . 86 |
| 9.2 | Procedures for Reporting Adverse Events | . 87 |
| 9.3 | Procedures for Reporting a Serious Adverse Event | . 87 |
| 9.4 | Procedures for Unmasking of Study Medication | . 88 |
| Adm | inistrative Items | . 88 |
| 10.1 | Protection of Human Subjects | . 89 |
| | 10.1.1 Compliance with Informed Consent Regulations (US 21 CFR Part 50) at Relevant Country Regulations | |
| | 10.1.2 Compliance With IRB or IEC Regulations | |
| | 10.1.3 Compliance With Good Clinical Practice | . 89 |
| | 10.1.4 Compliance With Electronic Records; Electronic Signatures Regulations (US 21 CFR Part 11) | |
| 10.2 | | |
| 10.4 | | |
| | 8.6<br>8.7<br>8.8<br>8.9<br>8.10<br>Advo<br>9.1<br>9.2<br>9.3<br>9.4<br>Adm<br>10.1 | 8.6 Unscheduled Visits |

| | | 10.4.1 Source Documents | 90 |
|---|---|---|---|
| | | 10.4.2 Case Report Form Completion. | 91 |
| | | 10.4.3 Study Summary | |
| | | 10.4.4 Retention of Documentation | 92 |
| | 10.5 | Labeling, Packaging, and Return or Disposal of Study Medications/Treatments | 92 |
| | | 10.5.1 Labeling/Packaging | |
| | | 10.5.2 Clinical Supply Inventory | |
| | | 10.5.3 Return or Disposal of Study Medications/Treatments and/or Supplies | |
| | | Monitoring by the Sponsor | |
| | | Handling of Biological Specimens. | |
| | 10.8 | Publications | 94 |
| | 10.9 | Coordinating Investigator | 94 |
| | 10.10 | Video Recording and Gonioscopic Photography | 94 |
| 11. | Refe | rences | 95 |
| 12. | Attac | hments | 98 |
| | 12.1 | Package Insert | 98 |
| | 12.2 | Glossary of Abbreviations | 99 |
| | 12.3 | Protocol Amendment Summary | 01 |
| | | 12.3.1 Amendment 1 | 101 |
| | | 12.3.2 Amendment 2 | 113 |
| | | List of Tables | |
| Tab | le 1 | Treatment Groups | 10 |
| | | | _ |
| | | | 6 |
| | | | _ |
| | | | 6 |
| | | | _ |
| | | | 6 |



# Protocol Summary

Study Compound: Bimatoprost sustained-release (SR) biodegradable implants containing preservative-free AGN-192024 (bimatoprost)

#### Phase: 3

## Study Objectives:

To evaluate the intraocular pressure (IOP)-lowering efficacy and safety of 2 dose strengths of Bimatoprost SR in patients with open-angle glaucoma (OAG) or ocular hypertension (OHT) after initial and repeated administrations

## Clinical Hypotheses:

At least 1 dose strength ( $10 \mu g$  or  $15 \mu g$ ) of Bimatoprost SR will have an IOP-lowering effect that is noninferior to that of topically administered timolol maleate 0.5% (hereafter referred to as timolol) eye drops in patients with OAG or OHT following single and repeat administration.

Bimatoprost SR administered intracamerally in dose strengths of 10  $\mu$ g or 15  $\mu$ g will have an acceptable safety profile in patients with OAG or OHT following single and repeat administration.

## Study Design

Structure: Phase 3, multicenter, randomized, masked, parallel-group comparison (2 dose strengths of Bimatoprost SR versus active control), repeat administration

Duration: Approximately 22 months, consisting of screening of up to 28 days before washout, washout period of up to 42 days before initial administration of study medication, 52-week treatment period, plus 8 months extended follow-up

Study Treatment Groups: Bimatoprost SR dose groups: 10 µg and 15 µg

Control: Timolol eye drops plus Sham needleless procedure (that involves touching the eye at the area of insertion with a needleless applicator).

Dosage/Dose Regimen: Patients will receive 1 of 2 dose strengths of Bimatoprost SR or Control treatment in the study eye on Day 1 (with repeat administration of the same dose strength or Sham at Week 16 and Week 32).

Bimatoprost SR-treated patients will receive intracameral administration of Bimatoprost SR in the study eye using a prefilled applicator. Timolol vehicle eye drops will be used twice daily (BID; in the morning and evening) to mask the treatment of patients receiving Bimatoprost SR in the study eye. The fellow eye will receive a Sham needleless procedure (hereafter called Sham administration or Sham administration procedure) plus topical timolol eye drops, BID. Control group patients will receive a Sham administration plus timolol in both eyes.

All patients will be masked to their treatment group. Treatment groups are shown in Table 1.

Table 1 Treatment Groups

| Treatment | Study Eye Treatment | Fellow Eye Treatment |
|---|---|---|
| Bimatoprost SR 10 μg | Dose strength: 10 μg | Sham administration procedure |
| | Eye drops: Vehicle BID | Eye drops: Timolol BID |
| Bimatoprost SR 15 μg | Dose strength: 15 μg | Sham administration procedure |
| | Eye drops: Vehicle BID | Eye drops: Timolol BID |
| Control | Sham administration procedure | Sham administration procedure |
| | Eye drops: Timolol BID | Eye drops: Timolol BID |

BID = twice daily

The patients will begin self-administration of the study-provided eye drops (vehicle or timolol) in both eyes, starting with the evening dose on the first administration (Bimatoprost SR or Sham administration) day visit. Patients will continue self-administration of the study-provided eye drops in the morning (08:00  $\pm$  1 hour) and in the evening (20:00  $\pm$  1 hour) approximately 12 hours apart throughout the study, with the exception of the morning of a subsequent visit, on which the morning eye drop administration will be performed at the study site.

Randomization/Stratification: Randomization to treatment groups will use a 1:1:1 ratio (Bimatoprost SR 10  $\mu$ g:Bimatoprost SR 15  $\mu$ g:Control). Randomization will be stratified by baseline study eye Hour 0 IOP ( $\leq$  25 mm Hg or > 25 mm Hg).

*Visit Schedule*: Patients who complete the entire study without receiving nonstudy IOP-lowering medication in both eyes will have a minimum of 25 visits and 6 phone calls.



Patients who have not received nonstudy IOP-lowering medication (prohibited prior to Week 52) in both eyes will receive a repeat administration of Bimatoprost SR (or Sham administration in Control group study eyes and all fellow eyes) at the Week 16 and Week 32 visits as indicated. Administration should not occur if the investigator believes that there are any safety concerns. Patients who have received nonstudy IOP-lowering medication in both eyes will be followed for at least 12 months following the last administration of Bimatoprost SR or Sham, at which time they may exit early at the investigator's discretion.

#### Study Population Characteristics

Number of Patients: Approximately 600 patients will be enrolled in the study.

Condition/Disease: Patients with OAG (primary OAG, pseudoexfoliative glaucoma, or pigmentary glaucoma) or OHT who require IOP-lowering medications in both eyes. The eye that meets the entry criteria will be selected as the study eye. If both eyes meet the entry criteria, the eye with the higher IOP at baseline Hour 0 will be selected as the study eye. If both eyes have the same IOP at Hour 0, then the right eye will be designated as the study eye.

Key Inclusion Criteria:

- •
- Diagnosis of either OAG (ie, primary, pseudoexfoliation, or pigmentary glaucoma) or OHT in each
  eye and both eyes require IOP-lowering treatment (Note: diagnosis does not have to be the same in
  both eyes)
- •



Key Exclusion Criteria:

- The following surgical history:
  - a. History or evidence of complicated cataract surgery in the study eye: eg, surgery resulting in complicated lens placement (such as anterior chamber intraocular lens implant [IOL], sulcus IOL, aphakia, etc) or intraoperative complications (such as a posterior capsular tear [with or without vitreous loss], substantial iris trauma, etc)

Note: history of uncomplicated cataract surgery is not an exclusion.

b. History of phakic IOL insertion for refractive error correction in the study eye



Response Measures

Efficacy: Intraocular pressure measured by Goldmann applanation tonometry



## General Statistical Methods and Types of Analyses:

The intent-to-treat population (ITT) is defined as all randomized patients and will be used for demographic and efficacy analyses. The per protocol (PP) population will consist of the subset of the ITT population with no protocol deviations affecting the primary efficacy analysis and will be used to confirm the primary efficacy analysis. A list of patients excluded from the PP population will be finalized prior to database lock. The safety population is defined as all patients who received study drug treatment and will be used for safety analyses. Analyses in the ITT population will be based on the treatment to which a patient was randomized, and analyses in both the PP and safety populations will be based on the actual treatment a patient received.

Continuous variables will be summarized by descriptive statistics including sample size, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized by frequency and percentage.

The primary efficacy variable is study eye time-matched IOP change from baseline. Mean IOP change from baseline will be compared between each Bimatoprost SR dose strength and timolol for each hour (Hours 0 and 2) using the ITT population. The comparisons at Week 12 will be considered the primary analysis.

Intraocular pressure change from baseline will be analyzed using a mixed-effects model repeated measures (MMRM) approach. The model will include IOP time-matched change from baseline as the response variable and treatment, timepoint (Hours 0 and 2 at each visit of Weeks 2, 6, and 12), treatment-by-timepoint interaction, and baseline IOP stratification as fixed effects. Unstructured covariance matrix will be used for repeated measures on the same patient; if the model with unstructured covariance matrix fails to converge, multiple imputation (MI) will be implemented before MMRM.

Within the framework of this model, the mean difference between each Bimatoprost SR dose strength and timolol (Bimatoprost SR minus timolol) and the corresponding 2-sided 95% confidence interval will be provided for each hour (Hours 0 and 2) at each visit. The formal noninferiority test will be performed at Week 12 for each Bimatoprost SR dose strength versus timolol using a noninferiority margin of 1.5 mm Hg. A gatekeeping procedure will be used to control the overall type I error rate at the 0.05 level for each hour at Week 12, testing Bimatoprost SR 15  $\mu$ g against timolol first and followed by the comparison between Bimatoprost SR 10  $\mu$ g and timolol. The test of Bimatoprost SR 10  $\mu$ g versus timolol for a given hour at Week 12 is valid only if the noninferiority of Bimatoprost SR 15  $\mu$ g to timolol is demonstrated for the same timepoint. Bimatoprost SR 15  $\mu$ g (or 10  $\mu$ g) will be declared noninferior to timolol if the upper limit of the 95% confidence interval is  $\leq$  1.5 mm Hg for both Hours 0 and 2 at Week 12.

For the United States Food and Drug Administration (US FDA), the primary efficacy variable will be the study eye IOP. The primary analysis will be based on Weeks 2, 6, and 12 using the ITT population. Specifically, the following analysis will be performed: IOP will be analyzed using an MMRM approach based on the same model as described for the primary efficacy analysis of time-matched IOP change from baseline. Within the framework of this model, the mean difference between each Bimatoprost SR dose strength and timolol group and the corresponding 95% confidence interval will be provided for each hour (Hours 0 and 2) and each visit (Weeks 2, 6, and 12). A gatekeeping procedure will be used to control the overall type I error rate at the 0.05 level for each timepoint, testing Bimatoprost SR 15  $\mu$ g against timolol first and followed by the comparison between Bimatoprost SR 10  $\mu$ g and timolol. The test for Bimatoprost SR 10  $\mu$ g versus timolol for a given hour at a visit is valid only if the noninferiority of Bimatoprost SR 15  $\mu$ g to timolol has been demonstrated for the given timepoint. Each Bimatoprost SR dose strength that shows noninferiority to timolol at all 6 timepoints with a 1.5 mm Hg margin (ie, the upper limit of the 95% confidence interval is  $\leq$  1.5 mm Hg) will be declared clinically noninferior to timolol if the upper limit of the 95% confidence interval is

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) and will be summarized for all events regardless of causality and for treatment-related adverse events. Ocular adverse events and safety variables will be tabulated by study eye and fellow eye within each treatment dose strength or group, and nonocular safety variables will be summarized by patient.

Sample Size Calculation: The sample size calculation is based on the primary efficacy analysis of the IOP for US FDA review because the sample size based on the primary efficacy analysis for other regions is expected to be smaller. Based on simulations, a sample size of 540 patients (180 per group) will provide approximately 95% and 81% power to show noninferiority (NI) of Bimatoprost SR 15  $\mu$ g and Bimatoprost SR 10  $\mu$ g, respectively, to timolol at all 6 scheduled timepoints based on an NI margin of 1.5 mm Hg and at 3 or more timepoints based on an NI margin of 1.0 mm Hg. Assuming a premature discontinuation rate of 10% within 12 weeks (before the primary database lock), approximately 600 patients (200 per group) are to be enrolled into this study.



15















# 1. Background and Clinical Rationale

#### 1.1 Glaucoma Overview

Glaucoma is a family of diseases commonly characterized by progressive optic neuropathy with associated visual field defects and is the leading cause of irreversible blindness in the world. Glaucoma is classified by Becker-Shaffer into 3 broad types: developmental, angle-closure, and open-angle glaucoma (OAG) (Stamper et al, 2009). Open-angle glaucoma is further categorized into primary OAG (POAG, sometimes also referred to as chronic OAG) and secondary OAG (which includes pigmentary and pseudoexfoliation glaucoma), the former being the predominant form of OAG. Primary OAG is characterized as a multifactorial optic neuropathy with a characteristic acquired atrophy of the optic nerve and loss of ganglion cells and their axons, developing in the presence of open anterior chamber (AC) angles, and manifesting characteristic visual field abnormalities (American Academy of Ophthalmology, 2010a). It is estimated that 2.25 million people in the United States (US) over the age of 40 years have POAG, half of whom are unaware of their disease despite demonstrable visual field loss (Quigley, 1996). Globally, over 60 million people are estimated to be affected by glaucoma (the majority of whom have open angle glaucoma) and these numbers are expected to increase over time (Quigley and Broman, 2006; Varma et al, 2011; Cook and Foster, 2012).

Although many risk factors have been associated with OAG elevated intraocular pressure (IOP) remains the most prominent factor and the only factor existing that ophthalmic intervention can reliably affect (Stamper et al., 2009). A number of controlled trials have demonstrated that lowering IOP will slow or delay the appearance or progression of glaucomatous damage. Large, randomized clinical trials such as the Ocular Hypertension Treatment Study (OHTS) (Kass et al. 2002) and the Early Manifest Glaucoma Trial (EMGT) (Heijl et al., 2002) addressed the value of early detection and lowering of elevated IOP in ocular hypertension (OHT) or POAG. The effects and parameters of various interventions in eyes with established glaucomatous damage were addressed by the Collaborative Initial Glaucoma Treatment Study (CIGTS) (Lichter et al, 2001) and the Advanced Glaucoma Intervention Study (AGIS) (AGIS, 2000). The currently available approaches to lowering IOP include pharmacological therapy, laser trabeculoplasty, incisional surgery, and cyclodestructive procedures. Each of these approaches has its own risk-benefit ratio. Because the risk-benefit ratio with drug therapy appears to be lower than that of surgical procedures, both historical and contemporary practice has been to attempt pharmacological treatment before resorting to other more invasive alternatives.

Patient nonadherence to topical therapy is one of the major challenges to preventing vision loss due to glaucoma, as consistent IOP reduction is associated with reduced risks of the development and progression of optic nerve damage (Friedman, 2009; Tsai, 2009). In patients that are nonadherent to medical therapy, guidelines are provided to clinicians for assisting patients with being adherent (Budenz, 2009). Nevertheless, frequently, patients with OAG or OHT not taking their medications will require incisional surgery to control the IOP. Some of the disadvantages of performing incisional surgery include the significant sight-threatening complications that can occur with surgery, such as the globe perforation, suprachoroidal hemorrhage, hypotony maculopathy, corneal decompensation, and cataract formation or progression that may occur with filtering surgery (Mosaed et al, 2009). Given the risks associated with incisional surgery, sustained-release formulations of ocular antihypertensive drugs are in development as an alternative to surgery for the management of elevated IOP (Knight and Lawrence, 2014).

# 1.2 Bimatoprost (LUMIGAN®)

Bimatoprost is a member of a series of unique prostanoid compounds that are potent and efficacious ocular antihypertensive agents (Woodward et al, 1994, 2001, and 2004). Bimatoprost appears to mimic the activity of biologically active prostamides (Study BIO-99-308; Matias et al, 2004). Chemically, prostamides differ from prostaglandin analogs by being neutral because they lack carboxylic acids (Krauss and Woodward, 2004). Prostamides can be biosynthetically derived from anandamide, an endogenous membrane lipid (Kozak et al, 2002; Weber et al, 2004; Woodward et al, 2001; Yu et al, 1997). The prostamide pathway leads to the biosynthesis of novel lipid amides that lower IOP.

The IOP-lowering efficacy of LUMIGAN (bimatoprost ophthalmic solution) 0.03% is well established. In phase 3 studies in patients with POAG or OHT, LUMIGAN administered once daily as monotherapy was superior to timolol at all timepoints (Higginbotham et al, 2002). This was further substantiated in the extension studies which followed patients in a masked manner for up to 4 years (Cohen et al, 2004; Williams et al, 2008; Study 192024-014). In clinical studies of patients with OAG or OHT with a mean baseline IOP of 26 mm Hg, the IOP-lowering effect of LUMIGAN once daily in the evening was 7 to 8 mm Hg (Cohen et al, 2004; LUMIGAN® Package Insert, 2012; Williams et al, 2008).

LUMIGAN was approved by the US Food and Drug Administration (FDA) in 2001.

Worldwide, LUMIGAN 0.03% is currently licensed and marketed in more than 80 countries and LUMIGAN 0.01% is licensed and marketed in more than 40 countries. Preservative-free

bimatoprost ophthalmic solution 0.03% has been approved since November 2012 for lowering IOP, and is currently marketed in 10 countries.

# 1.3 Bimatoprost SR

A sustained-release formulation of bimatoprost was developed at Allergan, Inc. to evaluate ocular antihypertensive therapies that do not require patient self-administration. Bimatoprost SR refers to the biodegradable, sustained-release, preservative-free bimatoprost implant which is preloaded in an applicator for administration, together they comprise the Bimatoprost Sustained Release product (and will henceforth be referred to as Bimatoprost SR). The Bimatoprost SR implant is injected into the AC via the corneal limbus using the prefilled applicator. The biodegradable polymer matrix gradually degrades to carbon dioxide and water so that there is no need to remove the Bimatoprost SR implant once the drug has been released. The Bimatoprost SR implant used in this study contains total preservative-free bimatoprost loads of 10 µg or 15 µg, to provide average daily release (as determined by in vitro studies) of approximately 110 ng or 170 ng, respectively, over an approximate 3-month duration in the AC. In contrast, a typical 35 μL drop of LUMIGAN 0.03% contains approximately 10 µg of bimatoprost. Thus, with topical therapy, a patient would have drug exposure to the ocular surface totaling approximately 900 μg over 3 months. Substantially reducing the total daily drug exposure to the eye and delivering the drug directly to the aqueous humor may reduce the adverse effects that occur with topical therapy. The Bimatoprost SR implant is expected to release drug over approximately 3 to 4 months, and > 75% polymer matrix degradation is expected within approximately 12 months. Although the biodegradation process of the Bimatoprost SR implant exceeds the drug release duration, experience from preclinical studies, the phase 1/2 clinical study 192024-041D, and approved intravitreal implants composed of similar biodegradable polymers provide support for the anticipated safety in a phase 3 clinical trial with repeated administration.

# 1.3.1 Nonclinical Studies with Bimatoprost SR

Pharmacology, toxicology, and pharmacokinetic studies with multiple dose strengths, implant sizes and formulations of Bimatoprost SR were done in 2 species (Beagle dog, Cynomolgus monkeys) with a range of anterior chamber angle sizes in order to support the clinical program. These studies build on the already considerable amount of nonclinical and clinical information available for topical bimatoprost (see Investigator's Brochure for additional details).



# 1.3.2 Other Biodegradable Ocular Implants

A number of sustained-release drug delivery implants using the Allergan biodegradable polylactic acid (PLA) and/or polylactic-co-glycolic acid (PLGA) NOVADUR® drug delivery system preceded the development of the Bimatoprost SR implant. The extensive clinical experience with previous intraocular implants demonstrates the safety and tolerability of an intraocular biodegradable implant administered into the eye via an applicator system. For example, late phase clinical trials of sustained-release implants have been completed for the OZURDEX® dexamethasone intravitreal implant using the NOVADUR drug delivery system for intraocular injections. Because Bimatoprost SR is similar to OZURDEX in a number of aspects and uses the NOVADUR drug delivery system for intraocular injections, these data may be supportive of the safety and tolerability of Bimatoprost SR in humans.

# 1.3.3 Clinical Study with Bimatoprost SR

Study 192024-041D was a Phase 1/2, paired-eye comparison evaluating the safety and efficacy of 4 dose strengths of Bimatoprost SR (6  $\mu$ g, 10  $\mu$ g, 15  $\mu$ g, or 20  $\mu$ g [2 × 10  $\mu$ g implants]), as single or repeat administration in one eye (study eye), versus the use of topical LUMIGAN® 0.03% in the fellow eye (nonstudy eye). The objective of this study was to evaluate the safety and IOP-lowering efficacy of Bimatoprost SR in patients with OAG.

A total of 109 patients received a single administration and 24 patients received a repeat administration of Bimatoprost SR. A trend in dose-response was observed across the 4 dose strengths that were tested. Data suggest that the implant may provide topical prostaglandin analog-like efficacy up to 3 to 4 months post-implantation in the majority of patients. Data following the second administration in the redosed patients showed similar IOP lowering to that observed following the first administration of Bimatoprost SR.

Bimatoprost SR showed an acceptable safety profile with single and repeat administrations in Study 192024-041D. Most adverse events were ocular, mild or moderate in severity, occurred within the first 2 days after Bimatoprost SR administration, and were considered related to the study drug administration procedure. There were no reports of serious study drug-related adverse events, and no new safety concerns were observed after the second treatment. Please refer to the Investigator's Brochure for details on reported safety findings.

# 1.4 Study Rationale

In the 192024-041D Phase 1/2 clinical study, results suggest that Bimatoprost SR provides IOP-lowering efficacy similar to topical prostaglandin analogs in the dose strengths proposed

for this Phase 3 investigation. Additionally, the safety profile of Bimatoprost SR at dose strengths of 20  $\mu$ g (2 × 10  $\mu$ g) or less in the Phase 1/2 study was acceptable, and supports additional clinical study in man. Study 192024-091 is a randomized, patient and efficacy evaluator-masked, parallel-group comparison to evaluate the safety and IOP-lowering effects of repeated administrations of 10  $\mu$ g or 15  $\mu$ g Bimatoprost SR in patients with OAG or OHT and open iridocorneal angles inferiorly in the study eye by clinical gonioscopy.

The 2 dose strengths of Bimatoprost SR will be compared versus a control group treated with the active comparator, topically applied timolol 0.5%. Timolol is a well-established treatment for IOP lowering in glaucoma and OHT, and has been used as a comparator in other IOP-lowering studies (Weinreb and Kaufman, 2009).

# Study Objectives and Clinical Hypotheses

# 2.1 Study Objectives

 To evaluate the IOP-lowering efficacy and safety of 2 dose strengths of Bimatoprost SR in patients with OAG or OHT after initial and repeated administrations

# 2.2 Clinical Hypotheses

- At least 1 dose strength (10 µg or 15 µg) of Bimatoprost SR will have an IOP-lowering effect that is noninferior to that of topically administered timolol maleate 0.5% (hereafter referred to as timolol) eye drops in patients with OAG or OHT following single and repeat administrations.
- Bimatoprost SR administered intracamerally in dose strengths of 10 µg or 15 µg will have an acceptable safety profile in patients with OAG or OHT, following single and repeat administrations.

# Study Design

This study is a multicenter, dose-ranging, randomized, parallel-group, patient and efficacy-evaluator masked 52-week evaluation (52-week treatment period with 8 months extended follow-up) of the safety and efficacy of Bimatoprost SR compared to timolol twice daily (BID) in patients with OAG or OHT. The patients and the evaluators of the primary endpoint (IOP) will be masked to the treatment received. The site coordinator and designated staff will not be masked to whether the patient received 1 of the two dose strengths of Bimatoprost SR or the Sham administration, but will be masked to the specific dose strength that the patient receives. Vehicle eye drops will be used BID to mask the treatment of

patients receiving Bimatoprost SR in the study eye. The fellow eye will receive a Sham administration plus topical timolol eye drops BID. Control group patients will receive a Sham administration plus timolol in both eyes (see Table 7). The study will be conducted at approximately 160 sites globally.

Two Bimatoprost SR dose strengths (10 µg or 15 µg) will be tested in this study. Patients will receive a scheduled second administration of Bimatoprost SR at 16 weeks following the first administration and a third scheduled administration at 16 weeks following the second administration (ie, 32 weeks after the initial administration). Control group patients will receive Sham administrations at all administration visits.

Table 7 Treatment Groups

| Treatment | Study Eye Treatment | Fellow Eye Treatment |
|---|---|---|
| Dimeterant CD 10 | Dose strength: 10 μg | Sham administration procedure |
| Bimatoprost SR 10 μg | Eye drops: Vehicle BID | Eye drops: Timolol BID |
| Dimeterant CD 15 | Dose strength: 15 μg | Sham administration procedure |
| Bimatoprost SR 15 μg | Eye drops: Vehicle BID | Eye drops: Timolol BID |
| Control | Sham administration procedure | Sham administration procedure |
| Control | Eyedrops: Timolol BID | Eyedrops: Timolol BID |

BID = twice daily

Patients will begin self-administration of the study-provided eye drops in both eyes starting with the evening dose on the first administration (Day 1) visit (at which they will receive Bimatoprost SR administration or Sham administration). Patients will continue self-administration of study-provided eye drops in the morning (at  $08:00 \pm 1$  hour) and in the evening (at  $20:00 \pm 1$  hour), which is approximately 12 hours apart. Patients will be instructed not to administer their drops on the morning of a study visit. Drops will be administered immediately after the Hour 0 IOP measurement.

The duration of the study for each patient is approximately 22 months (screening duration of up to 28 days before washout, plus washout of up to 42 days before the first administration, plus the 52-week treatment period, plus 8 months extended follow-up). Patients will be followed for at least 12 months after their last Bimatoprost SR (or Sham) administration, and may exit early at or after the twelfth month following the last administration if there are no safety concerns in the opinion of the investigator.

# 4. Study Population and Entry Criteria

## 4.1 Number of Patients

Enrollment of approximately 600 patients in total at approximately 160 sites, with approximately 200 patients per group, is planned to ensure 180 completed patients per group, assuming a premature discontinuation rate of 10%.

# 4.2 Study Population Characteristics

The study population consists of patients with OAG or OHT and an open iridocorneal angle inferiorly by clinical gonioscopy in the study eye, and OAG or OHT in the fellow eye, where both eyes require IOP-lowering medication. The eye that meets the entry criteria (Sections 4.3 and 4.4) will be selected as the study eye. If both eyes meet the entry criteria, the eye with the higher IOP at Baseline Hour 0 will be selected as the study eye. If both eyes have the same IOP, then the right eye will be designated as the study eye.

Angle qualification will be independently confirmed as being qualified by 2 ophthalmologists, and endothelial cell density qualification for study entry will be determined by the Reading Center based on specular microscopy assessment (see Protocol Procedure Manual for details).

## 4.2.1 Patients With Sickle Cell Trait or Disease

Patients with sickle cell trait or disease (or other hemoglobinopathies) may be enrolled at the discretion of the investigator based on an individual risk-benefit assessment. Because of a slightly higher risk of IOP elevation and intraocular complications in the setting of a microhyphema, patients with these disorders may undergo optional additional biomicroscopy and IOP measurements after injection/Sham injection at the investigator's discretion (see Section 8.4). Additional information about the Bimatoprost SR experience in patients with sickle trait is provided in the Investigator's Brochure.

## 4.3 Inclusion Criteria

The following are requirements for entry into the study:

- Male or female, ≥ 18 years of age
- 2. Written informed consent has been obtained

 Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable (eg, Written Authorization for Use and Release of Health and Research Study Information [US sites] and written Data Protection consent [EU sites])



Patient has the ability to understand and willingness to follow study instructions and is likely to complete all required visits and procedures

6.

 Diagnosis of either OAG (ie, primary, pseudoexfoliation, or pigmentary glaucoma) or OHT in each eye and both eyes require IOP-lowering treatment (Note: diagnosis does not have to be the same in both eyes)





# 4.4 Exclusion Criteria

The following are criteria for exclusion from participating in the study:

# Non-ocular Criteria for Exclusion

- Uncontrolled systemic disease
- Female patients who are pregnant, nursing, or planning a pregnancy, or who are of childbearing potential and not using a reliable means of contraception during the study (see Section 4.5.3)





- Any condition which would preclude the patient's ability to comply with study requirements, including completion of the study
- Patients who have a condition or are in a situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study



9. Previous enrollment in another Allergan Bimatoprost SR study



## Ocular Criteria for Exclusion



- 13. The following surgical history:
  - a. History or evidence of complicated cataract surgery in the study eye: eg, surgery resulting in complicated lens placement (such as anterior chamber intraocular lens implant [IOL], sulcus IOL, aphakia, etc) or intraoperative complications (such as a posterior capsular tear [with or without vitreous loss], substantial iris trauma, etc). Note: history of uncomplicated cataract surgery is not an exclusion.

14. Intraocular surgery (including cataract surgery) and/or any ocular laser surgery within the 6 months prior to treatment (Day 1) in the study eye




25. Anticipated need for any incisional or laser ocular surgery in either eye within the first 52 weeks of the study duration



28. Any history of trabeculectomy or other types of glaucoma surgery, including a glaucoma seton or aqueous bypass stents, in either eye



#### 4.5 Permissible and Prohibited Medications/Treatments

#### 4.5.1 Permissible Medications/Treatments

The fellow eyes of patients randomized to the Bimatoprost SR or Control groups will receive timolol BID for IOP lowering.

Intermittent use of artificial tear products is allowed if they are not taken  $\leq$  15 minutes before any study procedure or  $\leq$  15 minutes before or after topical administration of study medication. Intermittent use of ocular decongestants or antihistamines is allowed if not taken within 2 days prior to a scheduled visit and/or  $\leq$  15 minutes before or after topical administration of study medication. Use of artificial tear products and ocular decongestants or antihistamines may be restarted 3 days after any Bimatoprost SR (or Sham) administration procedure.

Use of postoperative topical ocular antibiotics, corticosteroids, and non-steroidal anti-inflammatory drugs (NSAIDs) from the Administration Day (on Day 1, Week 16, and Week 32) to Day 7 following administration is allowed.

Systemic beta-blocker containing medications are permitted, provided that the dose/dosing regimen has remained stable for at least 2 months prior to Screening, and is not anticipated to change during the duration of the study.

Required surgical procedures may be performed in the fellow eye only after completion of Week 52.

In addition, therapy considered necessary for the patient's welfare may be given at the discretion of the investigator. If concurrent medications may have an effect on study outcomes, these medications should be administered in dosages that remain constant throughout the entire duration of the study. If the permissibility of a specific medication/treatment is in question, please contact Allergan.

The use of systemic NSAIDs is also permitted.

In the unlikely event that the Bimatoprost SR implant requires removal for significant safety reasons, this may be performed at the discretion of the investigator following a discussion with the medical safety physician at Allergan (see Protocol Procedure Manual for details).

Note that in the event that the investigator performs an unanticipated incisional surgical procedure on the study eye during which ocular fluid is to be removed, ocular fluid/implant samples may be collected for analysis (see Protocol Procedure Manual for further details) at the investigator's discretion.

#### 4.5.2 Prohibited Medications/Treatments

The decision to administer a prohibited medication and/or treatment is done with the safety of the study participant as the primary consideration. When possible, Allergan should be notified before the prohibited medication/treatment is administered.

During the study, patients should not participate in other investigational drug or device studies.

#### Nonstudy IOP-lowering Medications

Use of any topical ophthalmic medication containing an ocular antihypertensive, other than use of study medication (timolol) in Control group or fellow eyes, is prohibited as concurrent therapy in either eye, unless necessary for the safety of the patient due to inadequate control of IOP as determined by the investigator. Inadequate control of IOP should be confirmed at a subsequent visit (scheduled or unscheduled visit). Prior to Week 52, the investigator will be expected to attest to the need for additional nonstudy IOP-lowering medication for safety reasons. After the Week 52 visit, nonstudy topical IOP-lowering medications will be permitted if in the investigator's clinical judgment the IOP is not adequately controlled at two consecutive visits. Initiation of medication in one eye should not automatically lead to initiation of medication in the other eye. Each eye should be evaluated on an individual basis when determining the need for additional nonstudy IOP-lowering medications. If nonstudy IOP-lowering medication is initiated prior to Week 52, the investigator will be expected to attest to the need for additional nonstudy IOP-lowering medication for safety reasons for each eye individually.

#### Contact Lenses

Use of soft contact lenses within 3 days and use of rigid gas permeable or hard contact lenses within 1 week prior to a scheduled study visit or Administration Day, or use of contact lenses of any kind within 1 week following any Bimatoprost SR (or Sham) administration in either eye is prohibited.

Contact lenses should be removed prior to instilling any study-provided eye drops and patients should wait at least 15 minutes before putting contact lenses back in the eyes after instilling topical drops.

#### Other Medications

The following medications (or classes of medications) and treatment procedures are not permitted as concurrent therapy during the study through 12 months after the last Bimatoprost SR or Sham administration <u>unless</u> the patient has already been treated with nonstudy IOP-lowering medication in <u>both</u> eyes:

 Subconjunctival, sub-Tenon's, intravitreal, or other ophthalmic injections of any medications in either eye

- Surgical procedures that are not related to Bimatoprost SR (or sham) administration procedures in the study eye (surgical procedures are allowed in the fellow eye after Week 52 as described in Section 4.5.1)
- Use of any topical ophthalmic medications (except as described above and in Section 4.5.1) in either eye.
- Use of any ophthalmic (including topical, intravitreal, sub-Tenon's, subconjunctival) corticosteroids in either eye from 2 months prior to the baseline visit through 12 months after the last administration, except for use of postoperative topical ocular coritcosteroids after administration as described in Section 4.5.1.
- Oral, intramuscular, or intravenous corticosteroids from 2 months prior to the baseline visit through the twelfth month after the last injection.
- Use of LATISSE<sup>®</sup> (bimatoprost for hypotrichosis) during the study period in either eye
- Systemic use of carbonic anhydrase inhibitors (eg, Diamox<sup>®</sup>)
- Any initiation of or alterations in systemic regimen of beta-blocker containing medications from 2 months prior to Screening through the final study visit

# 4.5.3 Definition of Females of (Non-)Childbearing Potential and/or Acceptable Contraceptive Methods

For purposes of this study, women will be considered of childbearing potential unless they are naturally postmenopausal or permanently sterilized (ie, hysterectomy). Natural menopause is defined as the permanent cessation of menstrual periods, determined retrospectively after a woman has experienced 12 months of amenorrhea without any other obvious pathological or physiological cause. For women of childbearing potential who may participate in the study, the following methods of contraception, if properly used, are generally considered reliable: hormonal contraceptives (ie, oral, patch, injection, implant), male condom with intravaginal spermicide, diaphragm or cervical cap with spermicide, vaginal contraceptive ring, intrauterine device, surgical sterilization (bilateral tubal ligation, bilateral salpingectomy), vasectomized partner, or true sexual abstinence (when this is in line with the preferred and usual lifestyle of the subject).

The investigator and each patient will determine the appropriate method of contraception for the patient during the participation in the study.

If a female becomes pregnant during the study, the investigator will notify the sponsor immediately after the pregnancy is confirmed and the patient will be exited from the study after appropriate safety follow-up. The investigator will (1) notify the patient's physician

that the patient was being treated with an investigational drug (unmask the study treatment as needed for pregnancy monitoring), and (2) follow the progress of the pregnancy. The investigator must document the outcome of the pregnancy and provide a copy of the documentation to Allergan.

#### Study Treatments

## 5.1 Study Treatments and Formulations

The clinical formulations of Bimatoprost SR contain preservative-free bimatoprost dispersed in a biodegradable polymer matrix (including PLA and PLGA). These biodegradable implants are preloaded in the applicator. The formulations used in this study are Bimatoprost SR 10 μg and Bimatoprost 15 μg.

#### 5.2 Control Treatments

For Sham administration, a needleless applicator is provided.

The following topical eye drops are also used as controls:

- Timolol 0.5% ophthalmic solution (maleate 0.68% (representing 0.5% timolol free base), benzalkonium chloride 0.01%, dibasic sodium phosphate heptahydrate, monobasic sodium phosphate, sodium hydroxide and/or hydrochloric acid to adjust pH, and purified water
- Timolol vehicle (
   timolol 0.5% ophthalmic solution and contains all ingredients of the above excluding timolol maleate

# 5.3 Methods for Masking

Patients in the Control group will receive timolol eye drops BID plus Sham administration in both eyes. Vehicle eye drops will be used BID to mask the treatment of patients receiving Bimatoprost SR in the study eye. Treatment for fellow eyes of patients assigned to 1 of the 2 Bimatoprost SR dose groups will be a Sham administration procedure + timolol eye drops BID.

The site coordinator and designated staff will not be masked to whether the patient received 1 of the 2 dose strengths of Bimatoprost SR or the Sham administration procedure, but will be masked to the specific implant dose strength. The patient and the remaining staff will be masked to the patient's treatment assignment. Efficacy IOP measurements will be masked by

using a 2-person reading method as described in Section 6.1.1 (for optional postoperative IOP measurements for patients with sickle cell disease or trait [or other hemoglobinopathies], see Section 8.4).

The site staff who perform IOP readings will be masked regarding the study eye (which eye received Bimatoprost SR or the Sham administration procedure), Bimatoprost SR dose strength, and the study treatments that are delivered in bottles. Site personnel and patients will be instructed and reminded throughout the study not to discuss study medication assignments to ensure maintenance of the masking.

Designated site personnel will be responsible for receiving, dispensing, and collecting study medication and performing drug accountability, as well as verification of patient dosing compliance; sites are encouraged to assign an unmasked staff member (eg, site coordinator) to this task to avoid unmasking additional personnel. Based on the randomization schedule, these designated personnel will dispense the study medication to the patient. All bottles will contain similar masked labels for the study, identifying the eye of administration by "Right" and "Left".

In the event that the patient requires topical corticosteroids or anti-inflammatory drops in only one eye during the 7 days after the administration procedure, in order to maintain masking the investigator will be instructed to dispense the required medication without disclosing which eye is the study eye, or the etiology of the signs/symptoms that require the medication.

The investigator is strongly encouraged not to use prohibited medications as outlined in Section 4.5.2. In order to maintain masking in the event that nonstudy IOP-lowering medications (prohibited prior to Week 52 unless required for a safety reason and attested to by the investigator) are administered, if a patient is started on a nonstudy IOP-lowering medication in only one eye, the patient will continue to use the study-provided eye drops in that eye as directed. The nonstudy IOP-lowering medication will be prescribed by the investigator according to local standard of care practices and used in addition to the study-provided eye drops in that eye. The eye not receiving a nonstudy IOP-lowering medication will continue to receive the study-provided eye drops as directed. If the eye receiving the nonstudy IOP-lowering medication is a Bimatoprost SR study eye, the eye will receive Sham administration on the administration day(s). If the eye receiving the nonstudy IOP-lowering medication is a Control group study eye or a fellow eye, the eye will continue to receive Sham administration on the administration day(s). If both eyes are receiving nonstudy IOP-lowering medications, the patient will discontinue use of the Allergan

study-provided eye drops and will not receive additional Bimatoprost SR or Sham administration (see Section 5.6.1). However, as described in Section 8.8, the patient will still remain in the study and be followed for 12 months following their last administration of Bimatoprost SR or Sham.

#### 5.4 Treatment Allocation Ratio and Stratification

Randomization to treatment groups will use a 1:1:1 ratio. Patients will be randomized to receive Bimatoprost SR (either 10  $\mu$ g or 15  $\mu$ g) plus vehicle eye drops, or a Sham administration procedure plus timolol eye drops, in the study eye. Randomization will be stratified by Baseline study eye Hour 0 IOP ( $\leq$  25 mm Hg or > 25 mm Hg).

## 5.5 Method for Assignment to Treatment Groups/Randomization

Prior to initiation of any study procedures, each patient who provides informed consent will be assigned a subject number that will serve as the patient's identification number on all study documents.

Eligible patients will be randomly assigned to 1 of 3 treatment groups in a 1:1:1 ratio to receive study Bimatoprost SR 10  $\mu$ g, Bimatoprost SR 15  $\mu$ g, or timolol. The randomization will be stratified by Baseline Hour 0 IOP (baseline study eye IOP  $\leq$  25 mm Hg or  $\geq$  25 mm Hg).

For determination of stratification group assignment for each patient, sites will be required to enter baseline IOP at Hour 0 data into electronic data capture (EDC). Electronic data capture will assign a stratification code associated with one of the stratification groups for the Baseline Hour 0 IOP.

At the time of randomization (Cycle 1 Day 1 Administration Day) an automated Interactive Voice/Web Response System (IV/WRS) will be used to manage the randomization and treatment assignment based on a randomization scheme prepared by Allergan Biostatistics. The site will enter the stratification group assignment code (obtained from the EDC) into IV/WRS at the time of randomization. A randomization number will be assigned to a patient according to the order of enrollment within each IOP stratum (baseline study eye Hour 0 IOP  $\leq$  25 mm Hg or  $\geq$  25 mm Hg) across the study. That is, IV/WRS will assign the next available randomization number to the patient at the time when the investigator requests randomization. Study medication will be labeled with medication kit numbers. The IV/WRS system will provide the site with the specific medication kit number(s) for each randomized patient at the time of randomization. Sites will dispense study medication according to the

IV/WRS instructions. Sites will also call the IVRS or log onto the IWRS at subsequent visits to obtain a study medication kit number for dispensing study medication. Sites will receive the IV/WRS confirmation notifications for each transaction. All notifications are to be maintained with the study source documents.

#### 5.6 Treatment Regimen and Dosing

The treatment groups are shown in Table 7. Patients randomized to 1 of the Bimatoprost SR dose groups will receive an intracameral administration of Bimatoprost SR in the study eye on Day 1, Week 16, and Week 32, in addition to using topical vehicle eye drops (1 drop BID). They will receive timolol eye drops (1 drop BID) plus Sham administration in the fellow eye. Patients randomized to the Control group will receive a Sham administration in both eyes on Day 1, Week 16, and Week 32, in addition to timolol eye drops (1 drop BID) in both eyes.

After the Administration Day 1 visit (Bimatoprost SR or Sham administration procedure), the patients should start administration of the study-provided eye drops in both eyes, starting with the evening dose. Patients should continue administering study-provided eye drops in the morning (at  $08:00 \pm 1$  hour) and in the evening ( $20:00 \pm 1$  hour), approximately 12 hours apart. Patients will be instructed <u>not</u> to administer the study-provided eye drops on the morning of study visits (except administration visits), and to bring their study medications to their visit for instillation immediately after the Hour 0 IOP measurements. If the patient arrives having taken the morning dose of study-provided eye drops, the site should attempt to reschedule within the visit window. Exception is made for the Day 2 study visit after any injection. As this visit is primarily for safety purposes, patients should undergo the visit regardless of whether they did or did not use the study medication that morning. Site personnel and patients will be reminded to take appropriate caution during administration of study medications during the visit to ensure maintenance of masking.

## 5.6.1 Treatment Regimen/Dosage Adjustments

Patients who have received nonstudy topical IOP-lowering medication (prohibited before Week 52 unless required for safety reasons due to inadequate IOP control and attested to by the investigator) in a Bimatoprost SR study eye will receive Sham administration in that eye on the Bimatoprost SR repeat administration day(s). Patients who have received nonstudy topical IOP-lowering medication in a fellow eye or a Control Group study eye will continue to receive Sham administration in that eye on the administration day(s).

Patients who have received nonstudy IOP-lowering medication in both eyes will not undergo Bimatoprost SR administration or Sham administration in either eye.

Patients who use nonstudy IOP-lowering medication (prohibited before Week 52 unless required for safety reasons due to inadequate IOP control and attested to by the investigator) in only one eye will be followed for the duration of the study. If used in both eyes, patients will be followed at minimum for 12 months after the last administration of Bimatoprost SR or Sham. Patients using nonstudy IOP-lowering medications in both eyes prior to the Week 16 or Week 32 Administration Day will not attend the administration visit(s), nor will they attend the Day 2, Days 4 and 8 (phone call), or 2-week visits (ie, Weeks 2, 18, and 34) following an administration. They would continue the schedule at Week 22 or Week 38, as appropriate for the administration cycle.

Patients who have received nonstudy IOP-lowering medication in both eyes before the time of the Month 14 visit are not required to attend the Month 14 or 18 visits unless the visit is 12 months after their last injection or Sham, at which time the patient may exit early and should complete all Month 20/Exit visit examinations. Patients who have received nonstudy IOP-lowering medication in both eyes by the time of the Month 16 visit are not required to attend the Month 18 visit, unless that visit is 12 months after their last injection or Sham, at which time the patient may exit early and should complete all Month 20/Exit visit examinations.

For patients who have not received nonstudy IOP-lowering medications by the time of study discontinuation or completion, poststudy evaluations regarding the need for IOP-lowering medications should be conducted according to the treating physician's clinical opinion.

# 5.7 Storage of Study Medications/Treatments

The study medication must be stored in a secure area and administered only to patients entered into the clinical study, at no cost to the patient, in accordance with the conditions specified in this protocol. Only assigned study personnel, authorized by the investigator, may have access to study medication. Bimatoprost SR and Sham needleless applicator must be stored in the original sealed foil pouch. Investigational medicinal product must be stored as described in the Investigator's Brochure. Sites must report any temperature excursions as described in the Protocol Procedure Manual or contact Allergan or its designee for further instructions.

For further details on storage, including requirements for study-provided eye drops, please refer to the Protocol Procedure Manual and/or contact Allergan.

## 5.8 Preparation of Study Medications/Treatments

Bimatoprost SR is loaded into the single use applicator during manufacturing and is provided within the applicator as a sterile, finished product. Study site personnel should notify Allergan or its designee immediately to advise of any situation in which the study medication is defective.

#### 5.9 Treatment Administration

Study medication must only be administered to patients who meet the eligibility criteria in accordance with the conditions specified in this protocol. Medication will be labeled with either a single panel label or booklet label. Records of use of medication kit numbers for each patient will be maintained by the site and recorded in the electronic case report form (eCRF) as appropriate.

## 5.9.1 Patient Preparation

Administration Day assessments (including vital signs and query for concomitant medications and adverse events) should be completed as outlined in Section 8.4. At least 3 administrations of a broad spectrum topical ophthalmic antibiotic drop and topical anesthetic drop should be administered to each eye approximately every 5 minutes beginning approximately 15 minutes prior to the procedure. With the patient in a supine position, the eye and conjunctival fornices should be irrigated with 5% ophthalmic povidone-iodine solution and the lids and surrounding orbital area should be prepped and draped according to the standard protocol detailed in the Protocol Procedure Manual.

## 5.9.2 Study Treatment Location

At the discretion of the investigator, Bimatoprost SR (or Sham) administration may be performed at an Ambulatory Surgical Center (ASC; free standing or hospital based) or in the office setting (eg, in a procedure room with an operating microscope). As a standard ASC technique an intravenous catheter may be placed and intravenous sedatives may be used at the discretion of the investigator and/or anesthesiologist. The Ambulatory Surgical Center may have standard operating procedures that require an electrocardiogram and/or a chest radiograph performed prior to the procedure. A separate standard consent to have the procedure at an Ambulatory Surgical Center may be required per the standard operating procedures at the facility.

Sterile technique will be practiced at all times.

## 5.9.3 Administration Technique

Intracameral administration of Bimatoprost SR must be performed by an ophthalmologist who has had adequate training and has been approved by Allergan to perform the procedure. The principal investigator at a site may designate a subinvestigator to perform the procedure, subject to Allergan approval and training. The study medication kit should be readily available during the procedure.

The procedure is described in detail in the Protocol Procedure Manual. In brief, following the sterile preparation and sterile field setup, an appropriately sized sterile lid speculum should be placed between the eyelids of the patient. The entrance site for the applicator needle is just anterior to the insertion of the conjunctiva through the clear cornea in the superior or temporal quadrant. The trajectory of the needle should be parallel to the iris plane. The eye is stabilized by either counter traction with a sterile toothed forceps or counter pressure with a cotton tipped applicator as the needle is advanced through the cornea. The actuator button is depressed until an audible and/or palpable click is heard. The Bimatoprost SR implant should be visible exiting the needle bevel into the aqueous humor. The needle is then immediately removed from the anterior chamber, and the wound is checked for aqueous leakage. Following removal of the lid speculum and sterile drape, additional drops of broad spectrum antibiotics should be applied.

The procedure for the second and third administrations of Bimatoprost SR is the same.

The procedure for all Sham administrations is the same; however, the Sham applicator will not have a needle and thus will not enter the anterior chamber (but should touch the eye at the area of recommended insertion).

#### 5.9.4 Immediate Posttreatment Observation

Following study treatment administration, the patient is allowed to sit upright and is kept for a minimum of 1 hour of observation. The surgeon will examine each of the patient's eyes to ensure that the anterior chamber is formed prior to the patient being released.

The patient will be supplied a bottle of topical ophthalmic antibiotic drops and instructions to use them for the next 3 days (including the day of the administration) in both eyes and to follow up as per protocol.

Prior to leaving the site, patients should be instructed to contact the study site immediately if they experience any adverse events after treatment. If the patient reports having experienced adverse events, these should be recorded on the appropriate eCRF.

The same posttreatment observation requirements apply after the second and third administrations of Bimatoprost SR or Sham administration.

Note: Patients with sickle cell disease or trait (or other hemoglobinopathies) may undergo optional biomicroscopy and IOP examination in both eyes 4 hours after each Bimatoprost SR administration (or Sham administration). This optional IOP examination is for postoperative purposes only, and as such does not require a masked, 2-person reading method. The IOP should be taken only once to avoid excessive postadministration (or Sham administration) manipulation of the eye, and should be taken by the investigator (or other unmasked, qualified personnel). This postadministration (or Sham administration) examination may be performed using a Goldmann applanation tonometer or a hand-held tonometer. (See the Study Procedure Manual for details.)

#### 5.10 Retreatment

Administration of Bimatoprost SR will occur at fixed intervals of 16 weeks, up to a total of 3 administrations. Patients will be readministered the Bimatoprost SR dose strength to which they were randomized unless in the investigator's opinion it would not be in the best interest of the patient to readminister Bimatoprost SR based on previous adverse events or safety concerns. Patients who have been treated with nonstudy IOP-lowering medication in only one eye will still attend administration visits; if the treated eye is the Bimatoprost SR study eye, the patient will receive a Sham administration in that eye. Control group study eyes and fellow eyes that have been treated with nonstudy IOP-lowering medications will continue to receive Sham administrations. Patients who have been treated with nonstudy IOP-lowering medication in both eyes will not attend the Administration Day visits, nor will they attend the Day 2, Days 4 and 8 (phone call), or the 2-week visits (ie, Weeks 2, 18, and 34) following an administration.

# 6. Response Measures and Summary of Data Collection Methods

Detailed information on equipment and methodology to be used is provided in the Protocol Procedure Manual.

# 6.1 Efficacy Measures

## 6.1.1 Primary Efficacy Measure

The primary efficacy measure, IOP, will be measured using a Goldmann applanation tonometer. Examiners masked to the treatment assignment should perform all efficacy IOP

measurements at approximately the same time of day for a given patient throughout the study whenever possible.

A 2-person reading method will be used for all efficacy IOP measurements, wherein 1 person adjusts the dial in a masked fashion and a second person reads and records the value. The right eye is to be measured first and the left eye measured second. Two consecutive measurements will be taken of each eye. If the first 2 measurements differ by > 1 mm Hg, a third measurement will be taken. If the first 2 measurements differ by 1 mm Hg or less, the IOP for the given eye will be the average of the 2 readings. If the difference between the first 2 measurements is > 1 mm Hg, the IOP for the given eye will be the median of the 3 readings.

All Hour 0 IOP examinations should be scheduled at  $08:00 \pm 1$  hour. As scheduling permits, the patient should have approximately the same Hour 0 time of day throughout the study. Hour 2 IOP examinations should occur 2 hours after the Hour 0 IOP exam. The acceptable window for the Hour 2 IOP examination is  $\pm$  30 minutes.

## 6.2 Safety Measures

The following will be collected and recorded on the appropriate eCRF page(s):

Adverse Events: All adverse events, from the moment the patient signs the informed consent form, will be monitored and recorded in the patient's source documents. All events will be reported to Allergan on an adverse event eCRF, including seriousness, severity, action taken and relationship to study drug. If adverse events occur, the first concern will be the safety of the study patient.

Weight and Height: Weight will be measured in pounds (lb) or kilograms (kg) using a scale. Height will be measured in inches (in) or centimeters (cm). Height and weight will be measured at screening as part of the demographic data; historical patient information and/or patient reports should not be used for either measurement.

Vital signs: Systolic and diastolic blood pressure and pulse rate will be measured after patients have been at rest (seated) for at least 5 minutes. Body temperature will be measured orally (or with an infrared forehead thermometer) and recorded as °F or °C.

Hematology, blood chemistry, and urinalysis: Blood and urine samples will be collected for blood chemistry and hematology panels and urinalysis.









## 6.4 Examination Procedures, Tests, Equipment, and Techniques

Study evaluations should be performed by the same investigator/subinvestigator throughout the study whenever possible. If it is not possible to use the same individual to follow the patient, then an attempt should be made to have investigators overlap (examine the patient together and discuss findings) for at least 1 visit.

# 6.4.1 Medical History, Physical Examination, and Vital Signs

# 6.4.1.1 Medical History

A standard medical history (including all relevant conditions that the patient has had in the past or currently has) will be captured in the patient source documents. All surgical procedures should have an associated medical history entry. Current medications as well as those stopped within 60 days prior to the screening visit and procedures within 90 days prior to the screening visit will be recorded. In addition, all previous medications taken for OAG

or OHT for at least 3 months prior to study entry will be recorded on the appropriate source document page.

## 6.4.1.2 Physical Examination

The patient will be examined by qualified medical personnel for any physical abnormality of the following systems: general appearance; head, eyes, ears, nose, and throat; heart/cardiovascular; lungs; abdomen; neurologic; extremities; back; musculoskeletal; lymphatic; and skin. The patient's height and weight will be recorded at the Screening visit only.

#### 6.4.1.3 Vital Signs

The below vital signs will be measured at all patient visits and should be recorded prior to any invasive procedures.

- Pulse rate (beats per minute [bpm]): the patient should be resting in a seated position for a minimum of 5 minutes prior to measurement. Pulse rate is then counted over 30 seconds (and multiplied by 2 to obtain bpm).
- Blood pressure (mm Hg): the patient should be resting in a seated position for a minimum of 5 minutes prior to measurement. Systolic/diastolic blood pressure will be measured with a sphygmomanometer (manual sphygmomanometer or automated blood pressure measuring device).
- Temperature (°C/°F): patients should be seated and the body temperature taken orally (or with an infrared forehead thermometer).

# 6.4.2 Pregnancy Testing

Urine will be collected from females of childbearing potential for pregnancy testing (urine pregnancy test). The urine test for pregnancy will be performed at the site utilizing the dipstick method at all specified timepoints. Serum testing may be performed instead of urine testing if required by the local institution.

## 6.4.3 Laboratory Procedures



Refer to the Central Laboratory Manual for further details regarding central laboratory collection and shipment procedures.

Laboratory test results will be forwarded from the central laboratory to the study site and to Allergan or its designee. The investigator or qualified site personnel must review all laboratory results for any adverse events. Laboratory test results that represent adverse events should be reflected on an adverse event eCRF page.

Evaluation and management of abnormal laboratory results should be conducted according to local site practice.

## 6.4.3.1 Hematology

Hematology will be measured and includes hematocrit, hemoglobin, glycated hemoglobin, (HbA1c), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), mean corpuscular volume (MCV), platelets, red blood cell (RBC) count, RBC morphology, total white blood cell (WBC) count and differential (neutrophils, bands, lymphocytes, monocytes, basophils, and eosinophils).

## 6.4.3.2 Serum Chemistry

Serum chemistry will include albumin, alkaline phosphatase, alanine transaminase (ALT), aspartate transaminase (AST), bicarbonate, calcium, chloride, creatinine, creatine kinase, direct bilirubin, glucose, indirect bilirubin, magnesium, phosphorous, potassium, sodium, total bilirubin, total cholesterol, total protein, urea nitrogen, and uric acid.

### 6.4.3.3 Urinalysis

Urine will be analyzed for clarity, color, bilirubin, blood, glucose, ketones, leukocyte esterase, nitrite, pH, protein, specific gravity, urobilinogen, and microscopic sediment (WBCs, RBCs, casts, bacteria, crystals, and epithelial cells).

# 6.5 Other Study Supplies

The following will be provided by Allergan or designated suppliers:

- All supplies needed for central laboratory blood and urine sampling (urinalysis, blood chemistry, and hematology), urine pregnancy test kits, and ocular fluid collection kits
- Shipping materials for shipment of laboratory samples to central laboratory
- Gonioscopy imaging equipment (selected sites only)

- As needed: AS-OCT, Specular Microscope, contact (ultrasound) pachymetry equipment, light meter, camera and related supplies for iris color photography
- Ancillary administration procedure supplies and postoperative topical ophthalmic antibiotics may be supplied

Sites that are not able to receive supplies from Allergan due to country regulations will need to provide their own supplies.

Allergan will not be providing any nonstudy IOP-lowering medications.

### 6.6 Summary of Methods of Data Collection

This study will use eCRFs using remote electronic data capture through a qualified third party vendor. The data will be entered on the eCRFs in a timely manner on an ongoing basis. The investigator is responsible for ensuring that data are properly recorded on each patient's eCRFs and related documents. An investigator who has signed the protocol signature page should personally sign for the case report forms (as indicated in the eCRFs) to ensure that the observations and findings are recorded on the eCRFs correctly and completely. A certified electronic copy of the eCRF including data corrections will be provided to the site for archiving at the end of the study.

A central laboratory

will be used for analysis of blood chemistry and hematology, urinalysis, and ocular fluid sample analysis (if ocular fluid is obtained). Laboratory data will be transferred to Allergan on a periodic basis throughout the study.

#### 7. Statistical Procedures

Three database locks are planned. The first database lock will take place after all patients have completed or prematurely discontinued before the Week 12 visit. Similarly, the database will be locked after all patients have completed or prematurely discontinued before Week 52 and Month 20/Exit. Analyses will be performed after each lock. Prior to the first database lock a detailed analysis plan will be finalized. To maintain the integrity of the ongoing study, Allergan study personnel who are directly involved in data handling and supporting the trial (such as the clinical study team) will remain masked to treatment assignment of individual patients during the study. To avoid potential data unmasking between locks and to protect trial integrity, study statistical personnel who have been unmasked after each lock will no longer be involved directly in any ongoing masked study conduct. Another statistician, who is still masked to study treatment, will assume these

responsibilities until the next lock. Unmasked data handling and appropriate data and results access will be specified prior to each lock.

Efficacy analyses specific for the US FDA (Division of Transplant and Ophthalmology Products) review are described in Section 7.6.

The details of all analyses will be provided in the analysis plan.

### 7.1 Analysis Populations

The intent-to-treat population (ITT) is defined as all randomized patients and will be used for demographic and efficacy analyses. The per protocol (PP) population will consist of the subset of the ITT population with no protocol deviations affecting the primary efficacy analysis and will be used to confirm the primary efficacy analysis. A list of patients excluded from the PP population will be finalized prior to database lock. The safety population is defined as all patients who received study drug treatment and will be used for safety analyses. Analyses in the ITT population will be based on the treatment to which a patient was randomized, and analyses in both PP and safety populations will be based on the actual treatment a patient received.

# 7.2 Collection and Derivation of Primary and Secondary Efficacy Assessments

The primary efficacy measurement is IOP, which will be measured in each eye using the Goldmann applanation tonometer. Two consecutive measurements will be taken for each eye. If these 2 measurements differ by > 1 mm Hg then a third measurement will be performed. If the first 2 measurements differ by 1 mm Hg or less, or a third measurement is required but only 2 measurements are obtained, then the IOP value for a given eye is the average of the 2 measurements. If 3 measurements are required (ie, the first 2 measurements differ by > 1 mm Hg) and obtained, then the IOP value for the given eye is the median of the 3 measurements. If, for any reason, only a single measurement is obtained, then this measurement will be used as the IOP value.

To avoid confounding of efficacy data, IOP measurements obtained after initiating the use of nonstudy IOP-lowering medication in an eye will be excluded from the calculation of the summary statistics and the statistical analyses for that eye but raw values will be presented in the listings.

## 7.2.1 Primary Efficacy Variable

The primary efficacy variable is the study eye time-matched IOP change from baseline (follow-up minus time-matched baseline) at each hour evaluated (Hours 0 and 2).

#### 7.2.2 Secondary Efficacy Variable

The secondary efficacy variable is time-matched IOP.

### 7.3 Hypothesis and Methods of Analysis

In general, continuous variables will be summarized by descriptive statistics including sample size, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized by frequency and percentage.

### 7.3.1 Primary Efficacy Analyses

The primary efficacy variable is the study eye time-matched IOP change from baseline. Mean IOP change will be compared between each Bimatoprost SR dose strength and the timolol group for each hour (Hours 0 and 2) using the ITT population. The comparisons at Week 12 will be considered the primary analysis.

The null and alternative hypotheses for the comparison between a given Bimatoprost SR dose strength and timolol at each hour of Week 12 are:

- Null hypothesis: the difference in mean IOP change from baseline between the given Bimatoprost SR dose strength and timolol (Bimatoprost SR minus timolol) is > 1.5 mm Hg.
- Alternative hypothesis: the difference (Bimatoprost SR minus timolol) in mean IOP change from baseline between the given Bimatoprost SR dose strength and timolol is ≤ 1.5 mm Hg.

Intraocular pressure change from baseline will be analyzed using a mixed-effects model repeated measures (MMRM) approach. The model will include IOP time-matched change from baseline as the response variable and treatment, timepoint (Hours 0 and 2 at each visit of Weeks 2, 6, and 12), treatment-by-timepoint interaction, and baseline IOP stratification as fixed effects. Unstructured covariance matrix will be used for repeated measures on the same patient; if the model with unstructured covariance matrix fails to converge, multiple imputation (MI) will be implemented before MMRM. The details of the model specifications will be provided in the analysis plan.

Within the framework of this model, the mean difference between each Bimatoprost SR dose strength and timolol (Bimatoprost SR minus timolol) and the corresponding 2-sided 95% confidence interval will be provided for each hour (Hours 0 and 2) at each visit. The formal noninferiority test will be performed at Week 12 for each Bimatoprost SR dose strength versus timolol using a noninferiority margin of 1.5 mm Hg. A gatekeeping procedure will be used to control the overall type I error rate at the 0.05 level for each hour at Week 12, testing Bimatoprost SR 15  $\mu$ g against timolol first and followed by the comparison between Bimatoprost SR 10  $\mu$ g and timolol. The test of Bimatoprost SR 10  $\mu$ g versus timolol for a given hour at Week 12 is valid only if the noninferiority of Bimatoprost SR 15  $\mu$ g to timolol is demonstrated for the same timepoint. Bimatoprost SR 15  $\mu$ g (or 10  $\mu$ g) will be declared noninferior to timolol if the upper limit of the 95% confidence interval is  $\leq$  1.5 mm Hg for both Hours 0 and 2 at Week 12.

Sensitivity analyses of handling missing data will be performed using multiple imputation.

## 7.3.2 Secondary Efficacy Analyses

Secondary efficacy analyses comparing each Bimatoprost SR dose strength and timolol to test the no-difference null hypothesis will be performed at scheduled visits (Weeks 2, 6, and 12) and hours for (1) IOP and (2) time-matched IOP change from baseline.

The analysis of time-matched IOP change from baseline utilizes the identical model as that described for the primary analysis in Section 7.3.1 with the same 2-sided 95% confidence intervals constructed at each hour and each visit for the mean difference between each Bimatoprost SR dose strength and timolol (Bimatoprost SR minus timolol). An upper 95% confidence limit of the mean difference that is less than zero corresponds to a significant difference in favor of the given Bimatoprost SR dose strength for the given timepoint.

Each Bimatoprost SR dose strength that demonstrates the following at all scheduled timepoints within the 12-week period (at Hours 0 and 2 at Weeks 2, 6, and 12) will be considered superior to timolol:

 The upper 95% confidence limit of the mean difference is less than zero (ie, a significant difference in favor of the given Bimatoprost SR dose strength)

The analysis of IOP will be similarly performed as described above with IOP replacing timematched IOP change from baseline in the analysis model.

58



## 7.3.4 Safety Analyses

The Medical Dictionary for Regulatory Activities (MedDRA) nomenclature will be used to code adverse events. Adverse events will be coded from the verbatim text into preferred term and system organ class (SOC). The number and percent of patients reporting treatment emergent adverse events will be tabulated based on the primary SOC and preferred terms. Summary tables will be generated for all adverse events regardless of causality as well as treatment-related adverse events for the entire study and by treatment cycle.



## 7.4 Subgroup Analyses

Subgroup analyses for the primary variable will be performed

# 7.5 Interim Analyses

No interim analysis is planned for this study. Each database lock will correspond to a milestone and statistical analysis when all randomized patients have either completed or exited from the targeted visit.

## 7.6 Analyses for US FDA

Primary Efficacy Analyses

For the US FDA review, the primary efficacy variable will be the study eye IOP. The primary analysis will be based on Weeks 2, 6, and 12 using the ITT population. Mean IOP will be compared between each Bimatoprost SR dose strength and timolol for each hour (Hours 0 and 2) at Weeks 2, 6, and 12.

The null and alternative hypotheses for the comparison between a given Bimatoprost SR dose strength and timolol for each hour at each visit are:

- The null hypothesis is that the difference in mean IOP between the given Bimatoprost SR dose strength and timolol (Bimatoprost SR minus timolol) is > 1.5 mm Hg.
- The alternative hypothesis is that the difference (Bimatoprost SR minus timolol) in mean IOP between the given Bimatoprost SR dose strength and timolol is ≤ 1.5 mm Hg.

IOP will be analyzed using an MMRM approach based on the same model as described in Section 7.3.1. Within the framework of this model, the mean difference between each Bimatoprost SR dose strength and timolol and the corresponding 2-sided 95% confidence interval will be provided for each hour (Hours 0 and 2) and each visit (Weeks 2, 6, and 12). A gatekeeping procedure will be used to control the overall type I error rate at the 0.05 level at each timepoint, testing Bimatoprost SR 15 μg against timolol first and followed by the comparison between Bimatoprost SR 10 μg and timolol. The test for Bimatoprost SR 10 μg versus timolol for a given hour at a visit is valid only if the noninferiority of Bimatoprost SR 15 μg to timolol has been demonstrated for the given timepoint.

Each Bimatoprost SR dose strength that shows noninferiority to timolol at all 6 timepoints with a 1.5 mm Hg margin (ie, the upper limit of the 95% confidence interval is  $\leq$  1.5 mm Hg) will be declared clinically noninferior to timolol if the upper limit of the 95% confidence interval is  $\leq$  1.0 mm Hg for 3 or more timepoints.

Sensitivity analyses of handling missing data will be performed using multiple imputation.

Secondary Efficacy Analyses

For each Bimatoprost SR dose strength which demonstrates efficacy (clinical noninferiority) as described in the primary efficacy analyses, secondary efficacy analyses comparing the Bimatoprost SR dose strength and timolol to test the no-difference null hypothesis will be

performed at scheduled visits (Weeks 2, 6, and 12) and hours for IOP. A gatekeeping procedure will be used to control the overall type I error rate at the 0.05 level within each dose strength; the specific sequence of the tests will be provided in the analysis plan.



## 7.7 Sample Size Calculation

The sample size calculation is based on the primary efficacy analysis of the IOP for US FDA review since the sample size based on the primary efficacy analysis for other regions is expected to be smaller.

The sample size is estimated based on a 2-sided t-test with  $\alpha$  = 0.05 at each timepoint and the assumption that the mean IOP difference between Bimatoprost SR 10  $\mu$ g and timolol is -0.25 mm Hg (ie, Bimatoprost SR 10  $\mu$ g is 0.25 mm Hg better in IOP-lowering than timolol) at Weeks 2 and 6 and 0 mm Hg at Week 12, with a common standard deviation of 4.0 mm Hg and a common within-subject correlation of 0.6. It is also assumed that the efficacy (IOP-lowering effect) of Bimatoprost SR 15  $\mu$ g is better than that of Bimatoprost SR 10  $\mu$ g by 0.25 mm Hg at each timepoint (Hours 0 and 2). These assumptions are based on the data obtained from the ongoing clinical study 192024-041D. Based on simulations, a sample size of 540 patients (180 per group) will provide approximately 95% and 81% power to show noninferiority (NI) of Bimatoprost SR 15  $\mu$ g and Bimatoprost SR 10  $\mu$ g, respectively, to timolol at all 6 scheduled timepoints based on an NI margin of 1.5 mm Hg and at 3 or more timepoints based on an NI margin of 1.0 mm Hg. Assuming a premature discontinuation rate of 10% within 12 weeks (before primary database lock), approximately 600 patients (200 per group) are to be enrolled into this study.

## 8. Study Visit Schedule and Procedures

Patients who complete the entire study without receiving nonstudy IOP-lowering medication will have a minimum of 25 visits and 6 phone calls.



### 8.1 Patient Entry Procedures

### 8.1.1 Overview of Entry Procedures

Prospective patients as defined by the criteria in Sections 4.3 and 4.4 (inclusion/exclusion criteria) will be considered for entry into this study.

## 8.1.2 Informed Consent and Patient Privacy

The study will be discussed with the patient and a patient wishing to participate must give informed consent prior to any study-related procedures or change in treatment. The patient must also give authorization (US only), data protection consent (Europe only), and other written documentation in accordance with the relevant country and local privacy requirements (where applicable) prior to any study-related procedures or change in treatment.

Each patient who provides informed consent will be assigned a subject number that will be used on patient documentation throughout the study.

#### 8.2 Washout Intervals

All patients must provide informed consent prior to beginning any drug washout for the purposes of inclusion in this study. Patients currently being treated with IOP-lowering medication(s) in either eye will begin washout of these medication(s) following completion of the screening procedures. The Screening and Washout periods may not be concurrent. The Washout period will be up to 42 days depending on the minimum washout period schedule below.

If patients cannot discontinue their prescribed therapy for up to 6 weeks to meet the washout period for study entry, the investigator may switch the patient's medication to one that requires a shorter washout interval during the washout of the original medication (Table 8). Nonetheless, the investigator should adhere to the minimum washout period for all IOP-lowering medications as indicated in Table 8.

If, after initial washout, the IOP does not meet entry criteria and the investigator believes this is due to inadequate washout, if time remains in the Washout period, he/she may perform additional washout, as long as the total Washout period does not exceed 42 days.



For patients undergoing a washout, interim safety evaluation(s) of IOP at some time during the washout period may be performed at the discretion of the investigator.

Note: Medications should only be discontinued (washed out) if the investigator feels that it is safe and appropriate, and if the patient is willing to discontinue the medication for the duration of the study. If the medication cannot be discontinued, then the patient will not be eligible for study entry.

## 8.3 Procedures for Final Study Entry

The results from the screening ocular and physical examinations, and laboratory tests (hematology/blood chemistry/urinalysis) must be evaluated and determined to be acceptable to the investigator prior to the patient's entry into the study. If repeat laboratory tests are done, the results must be reviewed prior to study treatment initiation on Day 1. Reading Center qualification of endothelial cell density must be confirmed by the Baseline visit. After confirmation of eligibility on Day 1, IV/WRS is contacted for randomization. However, this contact for randomization may take place at the end of the Baseline visit if needed. See Section 5.5 for the method for assignment to treatment groups/randomization.

A patient is considered to have enrolled in the study at the time of the first study treatment administration (or Sham).


























#### 8.5 Instructions for the Patients

Patients should be instructed to strictly follow the study visit schedule and to report all changes in their condition to the investigative site.

Instruction should be given to the patient to maintain a stable dose of any concomitant medication used chronically, or any new medications initiated during the study whenever possible. Patients should be instructed to communicate any changes to their medication at their next study visit. Patients should also be reminded to contact the study site if they are experiencing any difficulties during their study participation.

Patients should keep the study medication bottles in the original kit that was provided and return the bottles to the designated (unmasked) site staff. Patients should be instructed that bottles of provided medications should only be used for 28 days each.

Patients will be instructed not to administer the study-provided eye drops the morning of study visits (except Administration Day visits) and to bring their study medications to their visit for instillation immediately after the Hour 0 IOP measurements. Site personnel and patients will be reminded to take appropriate caution during administration of study medications during the visit to ensure maintenance of masking. Patients should instill their morning dose of study-provided eye drops on the day of the Administration Day visits.

Patients should be instructed to remove their contact lenses before instillation of any topical ophthalmic medication, and to keep contact lenses out for at least 15 minutes after instillation of eye drops.

#### 8.6 Unscheduled Visits

Additional examinations may be performed as necessary to ensure the safety and wellbeing of patients during the study period. Unscheduled visit eCRFs should be completed for each unscheduled visit. An assessment of any adverse event should be completed.

# 8.7 Compliance with Protocol

Patients must be able to adhere to the study visit schedule; appropriate inclusion, exclusion, and treatment criteria; permitted and prohibited medication criteria; and testing parameters as described in the protocol. At each study visit, patients will be asked if they have used their study-provided eye drops as instructed and whether they have used any concomitant medications/therapies or had any concurrent procedures since the previous visit.

Patients should be scheduled for study visits as closely to the day specified in the visit schedule as possible.

### 8.8 Early Discontinuation of Patients

Patients may voluntarily withdraw from the study at any time.

Patients who have received nonstudy IOP-lowering medication in only one eye will be followed for the duration of the study through the Month 20 visit.

Patients who have received nonstudy IOP-lowering medication in both eyes, or who do not complete an Administration Day visit, may discontinue the study 12 months after the last Bimatoprost SR or Sham administration at which time they should complete the Month 20/Exit visit procedures.

Notification of early patient discontinuation from the study and the reason for discontinuation will be made to the sponsor and will be clearly documented on the appropriate eCRF.

When patients exit before Month 20, the site should complete all procedures for the Month 20/Exit visit at the patient's last visit.

#### 8.9 Withdrawal Criteria

After the first administration (or Sham), failure to undergo an Administration Day visit does not indicate total withdrawal from the study. Patients who have received nonstudy IOP-lowering medication in only one eye will continue through the duration of the study. Patients who have received nonstudy IOP-lowering medication in both eyes, or patients who do not undergo Cycle 2 or 3 (or both) Administration Visits, will still be followed for 12 months after the last Bimatoprost SR or Sham administration for safety reasons. These patients are eligible for Early Discontinuation (Early Exit) as described in Section 8.8, above.

The investigator should consider withdrawing a patient from the study early if any of the following criteria are met:

- Patient develops (or has an exacerbation of) a medical condition that, in the opinion
  of the investigator, compromises the patient's ability to participate in the study
- Patient develops (or has an exacerbation of) a medical condition that, in the opinion
  of the investigator, compromises the patient's ability to participate in the study
- Patient is unwilling or unable to continue to comply with study procedures
- Patient is unwilling or unable to continue in the study

If a patient develops (or has an exacerbation of) a medical condition that, in the opinion of the investigator, would put the patient at an unacceptable medical risk by continuing study participation, the patient will be withdrawn from the study.

Whenever possible, the decision to withdraw a patient from the study or study treatment should be discussed with Allergan.

# 8.10 Study Termination

The study may be stopped at his/her study site at any time by the site investigator. Allergan may stop the study (and/or the study site) for any reason with appropriate notification.

#### Adverse Events

Adverse events occurring during the study will be recorded on an adverse event eCRF. If adverse events occur, the first concern will be the safety of the study participants.

#### 9.1 Definitions

#### 9.1.1 Adverse Event

An adverse event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. In addition, during the screening period, adverse events will be assessed regardless of the administration of a pharmaceutical product.

Note: Adverse events must be collected once informed consent has been obtained, regardless of whether or not the patient has been administered study drug.

Progression of treatment indication including new or worsening of anticipated clinical signs or symptoms, which are collected as clinical efficacy variables and assessed as unequivocally associated with the disease progression and /or lack of efficacy, should NOT be reported as adverse events unless the disease progression is greater than anticipated in the natural course of the disease.

Adverse events will be assessed, documented, and recorded in the CRF throughout the study (ie, after informed consent has been obtained). At each visit, the investigator will begin by querying for adverse events by asking each patient a general, nondirected question such as "How have you been feeling since the last visit?" Directed questioning and examination will then be done as appropriate. All reported adverse events will be documented on the appropriate case report form.

#### 9.1.2 Serious Adverse Event

A serious adverse event is any adverse event occurring at any dose that results in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. (See Section 9.3 for procedures for reporting a serious adverse event.)

Allergan considers all cancer adverse events as serious adverse events. In addition, Allergan considers any abortion (spontaneous or nonspontaneous) as a serious adverse event.

Preplanned surgeries or procedures for pre-existing, known medical conditions for which a patient requires hospitalization is not reportable as a serious adverse event.

Any preplanned surgery or procedure should be clearly documented in the site source documents by the medically qualified investigator at the time of the patient's entry into the study. If it has not been documented at the time of the patient's entry into the study, then it should be documented as a serious adverse event and reported to Allergan.

# 9.1.3 Severity

A clinical determination will be made of the intensity of an adverse event. The severity assessment for a clinical adverse event must be completed using the following definitions as guidelines:

Mild Awareness of sign or symptom, but easily tolerated.

Moderate Discomfort enough to cause interference with usual activity.

Severe Incapacitating with inability to work or do usual activity.

Not applicable In some cases, an adverse event may be an 'all or nothing' finding

which cannot be graded.

# 9.1.4 Relationship to Study Drug or Study Procedure

A determination will be made of the relationship (if any) between an adverse event and the study drug or study procedure, as applicable. A causal relationship is present if a

determination is made that there is a reasonable possibility that the adverse event may have been caused by the drug or study procedure.

If an adverse event is deemed related to study treatment, the investigator will be asked to further delineate whether the adverse event was related to the administration procedure (versus the study medication).

Note: A study procedure occurring during the Screening/Baseline period can include a washout of medication or introduction of a run-in medication or study required diagnostic procedure.

# 9.2 Procedures for Reporting Adverse Events

Any adverse event must be recorded on the appropriate case report form.

All adverse events that are drug-related and unexpected (not listed as treatment-related in the current Investigator's Brochure) must be reported to the governing Institutional Review Board/Independent Ethics Committee (IRB/IEC) as required by the IRB/IEC, local regulations, and the governing health authorities. Any adverse event that is marked "ongoing" at the exit visit must be followed up as appropriate.

# 9.3 Procedures for Reporting a Serious Adverse Event

Any serious adverse event occurring during the study period (beginning with informed consent) and for at least 4 months after the last dose of study drug must be immediately reported but no later than 24 hours after learning of a serious adverse event. Serious adverse events must be reported to Allergan (or Agent of Allergan) as listed on the Allergan Study Contacts Page and recorded on the serious adverse event form. All patients with a serious adverse event must be followed up and the outcomes reported. The investigator must supply the sponsor and the IRB/IEC with any additional requested information (eg, autopsy reports and discharge summaries).

In the event of a serious adverse event, the investigator must:

 Notify Allergan immediately <u>by fax or email</u> using the serious adverse event form (contact details can be found on page 1 of the serious adverse event form); phone numbers and relevant Allergan personnel contacts are also on the front page of protocol.

- Obtain and maintain in his/her files all pertinent medical records, information, and medical judgments from colleagues who assisted in the treatment and follow-up of the patient.
- 3. Provide Allergan with a complete, written description of the adverse event(s) on the serious adverse event form describing the event chronologically, including any treatment given (eg, medications administered, procedures performed) for the adverse event(s). Summarize relevant clinical information about the event: signs, symptoms, diagnosis, clinical course and relevant clinical laboratory tests, etc. Include any additional or alternative explanation(s) for the causality which includes a statement as to whether the event was or was not related to the use of the investigational drug.
- Promptly inform the governing IRB/IEC of the serious adverse event as required by the IRB/IEC, local regulations, and the governing health authorities.

# 9.4 Procedures for Unmasking of Study Medication

When necessary for the safety and proper treatment of the patient, the investigator can unmask the patient's treatment assignment to determine which treatment has been assigned and institute appropriate follow-up care. When possible, the sponsor (Allergan Medical Safety Physician) should be notified prior to unmasking study medication. The investigator should inform the sponsor (Allergan Medical Safety Physician) of the unmasking if there is no notification prior to the unmasking.

The treatment assignment for the patient can be determined by designated site personnel calling into the IVRS or IWRS system via password protected access. The reason for breaking the code must be recorded in the patient's source documents.

#### 10. Administrative Items

This protocol is to be conducted in accordance with the applicable Good Clinical Practice (GCP) regulations and guidelines, eg, the International Conference on Harmonisation (ICH) Guideline on GCP.

# 10.1 Protection of Human Subjects

# 10.1.1 Compliance with Informed Consent Regulations (US 21 CFR Part 50) and Relevant Country Regulations

Written informed consent is to be obtained from each patient prior to any study-related activities or procedures in the study, and/or from the patient's legally authorized representative. If the patient is under the legal age of consent, the consent form must be signed by the legally authorized representative in accordance with the relevant country and local regulatory requirements.

There are special situations in which oral informed consent may be taken. Approval to utilize oral consent procedures and instructions on how to properly obtain oral informed consent must be obtained from Allergan personnel.

# 10.1.2 Compliance With IRB or IEC Regulations

This study is to be conducted in accordance with IRB regulations (US 21 CFR Part 56.103) or applicable IEC regulations. The investigator must obtain approval from a properly constituted IRB/IEC prior to initiating the study and reapproval or review at least annually. Allergan is to be notified immediately if the responsible IRB/IEC has been disqualified or if proceedings leading to disqualification have begun. Copies of all IRB/IEC correspondence with the investigator should be provided to Allergan.

# 10.1.3 Compliance With Good Clinical Practice

This protocol is to be conducted in accordance with the applicable GCP regulations and guidelines.

# 10.1.4 Compliance With Electronic Records; Electronic Signatures Regulations (US 21 CFR Part 11)

This study is to be conducted in compliance with the regulations on electronic records and electronic signature.

# 10.2 Changes to the Protocol

The investigator must not implement any deviation from or changes of the protocol without approval by Allergan and prior review and documented approval/favorable opinion from the IRB/IEC of a protocol amendment, except where necessary to eliminate immediate hazards

to study patients, or when the changes involve only logistical or administrative aspects of the study (eg, change in monitors, change of telephone numbers).

### 10.3 Patient Confidentiality

A report of the results of this study may be published or sent to the appropriate health authorities in any country in which the study drug may ultimately be marketed, but the patient's name will not be disclosed in these documents. The patient's name may be disclosed to the Sponsor of the study, Allergan, or the governing health authorities or the FDA if they inspect the study records. Appropriate precautions will be taken to maintain confidentiality of medical records and personal information.

# 10.3.1 Patient Privacy

Written authorization (US sites only), data protection consent (European sites only), and other documentation in accordance with the relevant country and local privacy requirements (where applicable) is to be obtained from each patient prior to enrollment into the study, and/or from the patient's legally authorized representative in accordance with the applicable privacy requirements (eg, the Health Insurance Portability and Accountability Act Standards for Privacy of Individually Identifiable Health Information ("HIPAA"), European Union Data Protection Directive 95/46/EC ["EU Directive"]).

In accordance with HIPAA requirements, additional purposes of this study may include publishing of anonymous patient data from the study.

#### 10.4 Documentation

#### 10.4.1 Source Documents

Source documents may include a patient's medical records, hospital charts, clinic charts, the investigator's patient study files, as well as the results of diagnostic tests such as X-rays, laboratory tests, and electrocardiograms. The investigator's copy of the case report forms serves as part of the investigator's record of a patient's study-related data.

The following information should be entered into the patient's medical record:

- Patient's name
- Patient's contact information

- The date that the patient entered the study, patient number, and medication kit numbers
- The study title and/or the protocol number of the study and the name of Allergan
- A statement that informed consent was obtained (including the date). A statement that
  written authorization (US sites only), data protection consent (EU sites only), or other
  country and local patient privacy required documentation for this study has been
  obtained (including the date).
- Dates of all patient study visits
- All concurrent medications (List all prescription and nonprescription medications being taken at the time of enrollment. At each subsequent visit, changes to the list of medications and any concurrent procedures should be recorded.)
- Occurrence and status of any adverse events (including any procedure-related adverse events due to complications)
- The date the patient exited the study, and a notation as to whether the patient completed the study or reason for discontinuation
- The results of laboratory tests performed by the site (eg, blood chemistry and hematology, urinalysis, and pregnancy tests)
- Documentation of the patient's medical history
- Vital signs, physical examination findings
- IOP and ophthalmic examination findings
- Dates of Bimatoprost SR or Sham administration procedure
- Documentation of whether any procedure including study treatment administration was performed according to the protocol, noting any deviations (if applicable)
- Binocular color photographs, visual field print-outs, treatment video (if taken),
   AS-OCT and macular OCT print-outs

# 10.4.2 Case Report Form Completion

The investigator is responsible for ensuring that data are properly recorded on each patient's case report forms and related documents. An investigator who has signed the protocol signature page should personally sign for the case report forms (as indicated in the case report forms) to ensure that the observations and findings are recorded on the case report forms correctly and completely. The case report forms are to be submitted to Allergan in a timely manner at the completion of the study, or as otherwise specified by Allergan and will be maintained in a central data repository.

# 10.4.3 Study Summary

An investigator's summary will be provided to Allergan within a short time after the completion of the study, or as designated by Allergan. A summary is also to be provided to the responsible IRB/IEC.

#### 10.4.4 Retention of Documentation

All study related correspondence, patient records, consent forms, patient privacy documentation, records of the distribution and use of all investigational products, and copies of case report forms should be maintained on file.

For countries falling within the scope of the ICH guidelines, the sponsor-specific essential documents should be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents should be retained for a longer period, however, if required by the applicable regulatory requirement(s) or if needed by the sponsor.

In addition, for countries not falling within the scope of the ICH guidelines, local regulatory requirements should be followed regarding the retention of clinical study documentation.

Allergan requires that it be notified in writing if the investigator wishes to relinquish ownership of the data so that mutually agreed-upon arrangements can be made for transfer of ownership to a suitably qualified, responsible person.

# 10.5 Labeling, Packaging, and Return or Disposal of Study Medications/Treatments

# 10.5.1 Labeling/Packaging

Packaged and labeled study medication will be supplied by Allergan.

The assembled Bimatoprost SR (or Sham applicator) is individually packaged into a laminated foil pouch with desiccant and sealed. The entire foil pouch package is terminally sterilized. Each pouch will be placed into its own carton. The medication will be identified as an investigational product. The study number and medication kit number will be identified on the medication labels.

The study-provided eye drops (timolol or timolol vehicle) will be identified as an investigational product and provided in identically appearing bottles packed in cartons. Each carton will contain 2 identically appearing bottles, each of which will be labeled for the left or right eye. The study number and medication kit number will be identified on the medication labels and cartons.

The study medication contents are described in Sections 5.1 and 5.2.

Designated site personnel will be responsible for receiving, dispensing, and collecting study medications that are delivered in bottles and performing drug accountability.

# 10.5.2 Clinical Supply Inventory

The investigator must keep an accurate accounting of the number of investigational units received from Allergan, dispensed to the patients, the number of units returned to the investigator by the patient, and the number of units returned to Allergan during and at the completion of the study. A detailed inventory must be completed for the study medication. The study medication must be dispensed only by an appropriately qualified person to patients in the study. The medication is to be used in accordance with the protocol by patients who are under the direct supervision of an investigator.

# 10.5.3 Return or Disposal of Study Medications/Treatments and/or Supplies

All clinical study medications/treatments and/or supplies will be returned to Allergan or Allergan designee for destruction. Used applicators will be disposed of immediately in a sharps container.

Any malfunctioning applicators should be returned to Allergan or designee. Written instructions provided by Allergan should be followed when returning a malfunctioning applicator to Allergan or its representative.

# 10.6 Monitoring by the Sponsor

A representative of the sponsor will monitor the study on a periodic basis. The determination of the extent and nature of monitoring will be based on considerations such as the objective, purpose, design, complexity, blinding, size, and endpoints of the study.

Authorized representatives of Allergan or regulatory authority representatives will conduct on-site visits to review, audit and copy study-related documents. These representatives will meet with the investigator(s) and appropriate staff at mutually convenient times to discuss study-related data and questions.

# 10.7 Handling of Biological Specimens

Laboratory specimens for blood chemistry panel, hematology including complete blood count with differential, and urinallysis will be sent to a centralized clinical laboratory

with certification from a recognized accreditation agency (eg, College of American Pathology [CAP] or Clinical Laboratory Improvement Amendments [CLIA] certification) to be assayed using validated methods. All blood and urine samples will be stored at the centralized clinical laboratory following testing, and will be discarded after a time period indicated by Allergan. Allergan shall have full ownership rights to any biological specimens/samples derived from the study.

See the Laboratory Manual and the Protocol Procedure Manual for procedural details.

#### 10.8 Publications

Allergan, as the sponsor, has proprietary interest in this study. Authorship and manuscript composition will reflect joint cooperation between multiple investigators and sites and Allergan personnel. Authorship will be established prior to the writing of the manuscript. As this study involves multiple centers, no individual publications will be allowed prior to completion of the final report of the multicenter study except as agreed with Allergan.

### 10.9 Coordinating Investigator

A signatory Coordinating Investigator will be designated prior to the writing of the Clinical Study Report.

# 10.10 Video Recording and Gonioscopic Photography

In consenting patients, the procedure of administering the Bimatoprost SR and/or Sham Administration may be video recorded. The video recording will be made of the eye as viewed through an operating microscope. The video recordings may be used to review the study procedure and/or for general research, education, or informational purposes.

In consenting patients, goniophotographic images of the inferior iridocorneal angle may be obtained.

The patient's decision about whether to allow video recording or gonioscopic photography will not affect their eligibility for participation in the study.

#### 11. References

AGIS Investigators. The Advanced Glaucoma Intervention Study (AGIS): 7. The relationship between control of intraocular pressure and visual field deterioration. Am J Ophthalmol. 2000;130:429-440.

American Academy of Ophthalmology Glaucoma Panel. Preferred Practice Pattern® Guidelines. Primary open-angle glaucoma. San Francisco, CA: American Academy of Ophthalmology; 2010a. 27 p.

Budenz DL. A clinician's guide to the assessment and management of nonadherence in glaucoma. Ophthalmology. 2009;116:S43-S47.

Cohen JS, Gross RL, Cheetham JK, VanDenburgh AM, Bernstein P, Whitcup SM. Two-year double-masked comparison of bimatoprost with timolol in patients with glaucoma or ocular hypertension. Surv Ophthalmol. 2004;49 (Suppl 1):S45-S52.

Cook C, Foster P. Epidemiology of glaucoma: What's new? Can J Ophthalmol. 2012;47:223-226.

Friedman DS. Introduction: new insights on enhancing adherence to topical glaucoma medications. Ophthalmology. 2009;116:S29.

Heijl A, Leske MC, Bengtsson B, Hyman L, Bengtsson B, Hussein M. Reduction of intraocular pressure and glaucoma progression: results from the Early Manifest Glaucoma Trial. Arch Ophthalmol. 2002;120:1268-1279.

Higginbotham EJ, Schuman JS, Goldberg I, Gross RL, VanDenburgh AM, Chen K, et al. One-year, randomized study comparing bimatoprost and timolol in glaucoma and ocular hypertension. Arch Ophthalmol. 2002;120:1286-1293.

Kass MA, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, et al. The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002;120:701-713.

Knight O'RJ, Lawrence SD. Sustained drug delivery in glaucoma. Current Opinion in Ophthalmology 2014;25(2):112-117.

Kozak KR, Crews BC, Morrow JD, Wang L-H, Ma YH, Weinander R, et al. Metabolism of the endocannabinoids, 2-arachidonylglycerol and anandamide, into prostaglandin, thromboxane, and prostacyclin glycerol esters and ethanolamides. J Biol Chem. 2002;277:44877-44885.

Krauss AH, Woodward DF. Update on the mechanism of action of bimatoprost: a review and discussion of new evidence. Surv Ophthalmol. 2004;49(Suppl 1):S5-11.

Lichter PR, Musch DC, Gillespie BW, Guire KE, Janz NK, Wren PA, et al. Interim clinical outcomes in the Collaborative Initial Glaucoma Treatment Study comparing initial treatment randomized to medications or surgery. Ophthalmology. 2001;108:1943-1953.

LUMIGAN® [Package Insert]. Irvine, CA: Allergan, Inc. 2012.

Matias I, Chen J, De Petrocellis L, Bisogno T, Ligresti A, Fezza F, et al. Prostaglandin ethanolamides (prostamides): in vitro pharmacology and metabolism. J Pharmacol Exp Ther. 2004;309:745-757.

Mosaed S, Dustin L, Minckler DS. Comparative outcomes between newer and older surgeries for glaucoma. Trans Am Ophthalmol Soc. 2009;107:127-33.

Quigley HA. Number of people with glaucoma worldwide. Br J Ophthalmol. 1996;80:389-393.

Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006;90:262-267. Doi: 10.1136/bjo.2005.081224. Downloaded from bjo.bm.com, April 9, 2014.

Stamper RL, Lieberman MF, Drake MV, eds. Introduction and Classification of the Glaucomas. In: Stamper RL, Lieberman MF, Drake MV, editors. Becker-Shaffer's Diagnosis and Therapy of the Glaucomas, 8th ed. Amsterdam, Netherlands: Mosby Elsevier; 2009;Chap 1:1-7.

Tsai JC. A comprehensive perspective on patient adherence to topical glaucoma therapy. Ophthalmology. 2009;116:S30-S36.

Varma R, Lee PP, Goldberg I, Kotak S. An assessment of the health and economic burdens of glaucoma. Am J Ophthalmol. 2011;152:515-522.

Weber A, Ni J, Ling KH, Acheampong A, Tang-Liu DD, Burk R, et al. Formation of prostamides from anandamide in FAAH knockout mice analyzed by HPLC with tandem mass spectrometry. J Lipid Res. 2004;45:757-763.

Weinreb RN, Kaufman PL. The Glaucoma Research Community and FDA look to the future: a report from the NEI/FDA CDER Glaucoma Clinical Trial Design and Endpoints Symposium. Inv Ophthalomol & Vis Sci. 2009;50(4):1497-1505.

Williams RD, Cohen JS, Gross RL, Liu CC, Safyan E, Batoosingh AL. Long-term efficacy and safety of bimatoprost for intraocular pressure lowering in glaucoma and ocular hypertension: year 4. Br J Ophthalmol. 2008;92:1387-1392.

Woodward DF, Chan MF, Burke JA, Cheng-Bennett A, Chen G, Fairbairn CE, et al. Studies on the ocular hypotensive effects of prostaglandin F2 alpha ester prodrugs and receptor selective prostaglandin analogs. J Ocul Pharmacol. 1994;10:177-193.

Woodward DF, Krauss AH, Chen J, Lai RK, Spada CS, Burk RM. The pharmacology of bimatoprost (Lumigan). Surv Ophthalmol. 2001;45(Suppl 4):S337-S345.

Woodward DF, Phelps RL, Krauss AH, Weber A, Short B, Chen J, et al. Bimatoprost: A novel antiglaucoma agent. Cardiovasc Drug Rev. 2004;22:103-120.

Yu M, Ives D, Ramesha CS. Synthesis of prostaglandin E2 ethanolamide from anandamide by cyclooxygenase-2. J Biol Chem. 1997;272:21181-21186.

# 12. Attachments

# 12.1 Package Insert

The appropriate package insert or Summary of Product Characteristics will be supplied to investigators in countries where timolol (study-provided eye drops) is marketed.

# 12.2 Glossary of Abbreviations

Term/Abbreviation Definition

ABMD Anterior Basement Membrane Disease

AC Anterior chamber

ARMD Age-related Macular Degeneration

ASC Ambulatory Surgical Center

AS-OCT Anterior segment optical coherence tomography

BCVA Best-corrected visual acuity

BID Twice daily

BLQ Below the limit of quantitation

CRF Case report form

DMEK Descemet's Membrane Endothelial Keratoplasty
DSEK Descemet's Stripping Endothelial Keratoplasty

eCRF Electronic case report form
EDC Electronic data capture

EU European Union

FDA Food and Drug Administration

GCP Good Clinical Practices
GLP Good Laboratory Practice

HIPAA Health Insurance Portability and Accountability Act

ICH International Conference on Harmonisation

IEC Independent Ethics Committee

IOL Intraocular lens implant
IOP Intraocular pressure

IRB Institutional Review Board

ITT Intent-to-treat

IV/WRS Interactive voice/web response system

MedDRA Medical Dictionary for Regulatory Activities

MMRM Mixed-effects model repeated measures

NI Noninferiority

NSAID Non-steroidal anti-inflammatory drug

OAG Open-angle glaucoma

OCT Optical coherence tomography

OHT Ocular hypertension

OU Both eyes

#### Term/Abbreviation Definition

PAS Peripheral anterior synechiae

PLA Polylactic acid

PLGA Polylactic-co-glycolic acid POAG Primary open-angle glaucoma

PP Per protocol
RBC Red blood cell

SC/T Patients with sickle cell disease or trait or other

hemoglobinopathies

SOC System Organ Class (MedDRA)

SR Sustained release
US United States
WBC White blood cell

# 12.3 Protocol Amendment Summary

#### 12.3.1 Amendment 1

Title: The Efficacy and Safety of Bimatoprost SR in Patients With Open-angle Glaucoma or Ocular Hypertension

Protocol 192024-091 Amendment 1

Date of Amendment: August 2015

#### Amendment Summary

This summary includes changes made to Protocol 192024-091 (approved September 2014). This protocol was amended to clarify some sections and to modify the inclusion/exclusion criteria.

Following is a summary of content-oriented changes that were made to each section of the protocol, and a brief rationale for these changes. Minor editorial and document formatting revisions have not been summarized.











| Section | Revision | Rationale |
|---|---|---|
| Section<br>4.5.1 | Revised the following: Intermittent use of ocular decongestants or antihistamines is allowed if not taken within 2 weeks days prior to a scheduled visit and/or ≤ 15 minutes before or after topical administration of study | Decreased to 2 days in order to reduce limitations on patients in a 2-year study. |
| | medication. Added the following: Required surgical procedures may be performed in the fellow eye only after completion of Week 52. | Because this is not a paired eye comparison, the fellow eye may have required surgery after the treatment period has been completed. |
| | Updated as follows: Note that in the event that the investigator performs an unanticipated incisional surgical procedure on the study eye during which ocular fluid is to be removed, ocular fluid/implant samples may be collected for analysis (see Protocol Procedure Manual for further details)—) at the investigator's discretion. | Revised the description of ocular fluid collection for clarity. |
| Section<br>4.5.2 | Nonstudy IOP-lowering Medications Use of any topical ophthalmic medication containing an ocular antihypertensive, other than use of study medication (timolol) in Control group or fellow eyes, is prohibited as concurrent therapy in either eye during the study through Week 52, unless necessary for the safety of the patient due to inadequate control of IOP as determined by the investigator. NonstudyInadequate control of IOP should be confirmed at a subsequent visit (scheduled or unscheduled visit). Prior to Week 52 the investigator will be expected to attest to the need for additional nonstudy IOP-lowering medication for safety reasons. After the Week 52 visit, nonstudy topical IOP-lowering medications will be permitted after the Week 52 visit, if in the investigator's clinical judgment the IOP is not adequately controlled at two consecutive visits at least 1 week apart. Initiation of medication in one eye should not automatically lead to initiation of medication in the other eye. Each eye should be evaluated on an individual basis when determining the need for additional non-study IOP-lowering medications. If nonstudy IOP lowering medication for week 52, the investigator will be expected to attest to the need for additional non-study IOP-lowering medication for | Updated text for clarity. |
| | Contact Lenses Use of soft contact lenses within 3 days and use of rigid gas permeable or hard contact lenses within 1 week prior to a scheduled study visit or Administration Day, or use of contact lenses of any kind within 1 week following any Bimatoprost SR (or Sham) administration in either eye is prohibited. | Updated text for clarity and to reduce limitations for patients who use contact lenses. |
| | Contact lenses should be removed prior to instilling any study-provided eye drops and patients should wait at least 15 minutes before putting contact lenses back in the eyes | |
| Section | Revision | Rationale |
|---|---|---|
| | after instilling topical drops. | |
| | Other Medications | |
| | <ul> <li>Surgical procedures that are not related to Bimatoprost</li> </ul> | |
| | SR (or sham) administration procedures in either eye | |
| | the study eye. (Surgical procedures are allowed in the | |
| | fellow eye after Week 52 as described in Section 4.5.1) | |
| | Use of any nonstudy topical ophthalmic medications | |
| | (except as described above and in Section 4.5.1) in | |
| | either eye | |
| | Use of soft contact lenses within 1 week and use of | |
| | rigid gase permeable or hard contact lenses within 2 | |
| | weeks prior to a scheduled study visit, or use of contact | |
| | lenses of any kind within 2 weeks following any | |
| | Bimatroprost SR (or Sham) administration in either eye | |
| Section<br>4.5.3 | For women of childbearing potential who may participate in the study, the following methods of contraception, if properly used, are generally considered reliable: hormonal contraceptives (ie, oral, patch, injection, implant), male condom with intravaginal spermicide, diaphragm or cervical cap with spermicide, vaginal contraceptive ring, intrauterine device, surgical sterilization (bilateral tubal ligation, bilateral salpingectomy), vasectomized partner, or true sexual abstinence, when this is in line with the preferred and usual lifestyle of the subject. | Updated text for clarity. |
| | The investigator will (1) notify the patient's physician that the patient was being treated with an investigational drug (Bimatoprost SR unmask the study treatment as needed for pregnancy monitoring), and (2) follow the progress of the pregnancy. | |

| Section | Revision | Rationale |
|---|---|---|
| Section 5.3 | The investigator is strongly encouraged not to use prohibited medications as outlined in Section 4.5.2. In order to maintain masking in the event that nonstudy IOP-lowering medications (prohibited prior to Week 52 unless required for a safety reason and attested to by the investigator) are administered, if a patient is started on a nonstudy IOP-lowering medication in only one eye, the patient will continue to use the study-provided eye drops in that eye as directed. The nonstudy IOP-lowering medication will be prescribed by the investigator according to local standard of care practices, and used in addition to the study-provided eye drops in that eye. The eye not receiving a nonstudy IOP-lowering medication will continue to receive the study-provided eye drops as directed. If the eye receiving the nonstudy IOP-lowering medication is a Bimatoprost SR study eye, the eye will receive Sham administration on the administration day(s). If the eye receiving the nonstudy IOP-lowering medication is a Control group study eye or a fellow eye, the eye will continue to receive Sham administration on the administration day(s). If both eyes are receiving nonstudy IOP-lowering medications, the patient will discontinue use of the Allergan study-provided eye drops and will not receive additional Bimatoprost SR or Sham administration (see Section 5.6.1).) However, as described in Section 8.8, the patient will still remain in the study and be followed for 12 months following their last administration of Bimatoprost SR or Sham. | Updated text for clarity. Updated text for clarity. |
| Section<br>5.6 | If the patient arrives having taken the morning dose of study-provided eye drops, the site should attempt to reschedule within the visit window. Exception is made for the Day 2 study visit after any injection. As this visit is primarily for safety purposes, patients should undergo the visit regardless of whether they did or did not use the study medication that morning.) | opales text for clarity. |
| Section<br>5.6.1 | Patients who have received nonstudy topical IOP- lowering medication (prohibited before Week 52 <u>unless required for safety reasons due to inadequate IOP control and attested to by the investigator)</u> in a Bimatoprost SR study eye will receive Sham administration in that eye on the Bimatoprost SR repeat administration day(s). Patients who use nonstudy IOP-lowering medication (prohibited before Week 52 <u>unless required for safety reasons due to inadequate IOP control and attested to by the investigator)</u> in only one eye will be followed for the duration of the study. | Updated text for clarity. |
| | Patients who have received nonstudy IOP-lowering medication in both eyes before the time of the Month 14 visit are not required to attend the Month 14 or 18 visits unless the visit is 12 months after their last injection or | Months 14 and 18 visits will be optional for patients already treated with nonstudy IOP-lowering medication in both eyes. |





| Section | Revision | Rationale |
|---|---|---|
| Sections<br>8.4.4.1<br>and<br>8.4.4.3 | | |
| Section<br>8.4.4.2 | | |
| Section<br>8.5 | Patients should be instructed to remove their contact lenses before instillation of any study-provided topical ophthalmic medication, and to keep contact lenses out for at least 15 minutes after instillation of eye drops. | Added information included in the patient drops instruction handout for consistency. |
| Section<br>8.8 | Patients who have received nonstudy IOP-lowering medication in both eyes, or who do not complete an Administration Day visit, may discontinue the study 12 months after the last Bimatoprost SR or Sham administration- at which time they should complete the Month 20/Exit visit procedures. | Updated text for clarity. |
| Section<br>8.9 | After the first administration (or Sham), failure to undergo an Administration visit does not indicate total withdrawal from the study. Patients who have received nonstudy IOP-lowering medication in only one eye will be followed for the duration of the study. Patients who have received nonstudy IOP-lowering medication in both eyes, or patients who do not undergo Cycle 2 or 3 (or both) administrations (or Sham administrations), will still be followed for 12 months after the last Bimatoprost SR or Sham administration for safety reasons. These patients are eligible for Early Discontinuation (Early Exit) as described in Section 8.8, above. •Patient develops (or has an exacerbation of) a medical condition that, in the opinion of the investigator, would | Updated text for clarity, as in this study design, patients are followed for 12 months after their last injection (or Sham) for safety purposes, and cessation of injection does not constitute study withdrawal. |
| | putcompromises the patient at an unacceptable medical risk by continuing patient's ability to participate in the study participation | |
| | If a patient develops (or has an exacerbation of) a medical condition that, in the opinion of the investigator, would put the patient at an unacceptable medical risk by continuing study participation, the patient will be withdrawn from the study. | |

#### 12.3.2 Amendment 2

Title: The Efficacy and Safety of Bimatoprost SR in Patients With Open-angle Glaucoma or Ocular Hypertension

Protocol 192024-091 Amendment 2

Date of Amendment: March 2017

#### Amendment Summary

This summary includes changes made to Protocol 192024-091 Amendment 1 (approved August 2015). This protocol was amended to change the screening requirement for angle eligibility confirmation in the study eye, modify/clarify the inclusion/exclusion criteria, clarify the statistical analyses, and change additional procedures for patients with sickle cell disease from required to optional.

Following is a summary of content-oriented changes that were made to each section of the protocol, and a brief rationale for these changes. Minor editorial and document formatting revisions have not been summarized.

## Section Revision Rationale Protoco1 Removed text from the visit schedule section referring to Updated to reflect changes in the Summary reading center confirmation of iridocorneal angle: body of the protocol. Screening (up to 28 days); Washout period of up to 42 days for both eyes (which may begin once screening procedures have been completed and the site has obtained confirmation of anterior segment optical coherence tomography [AS OCT] iridocorneal angle qualification from the Reading Center); Baseline (Days 3 to 1 up to 3 days) Updated the following key inclusion criteria: Updated the following key exclusion criterion: The following surgical history: a. History or evidence of complicated cataract surgery in the study eye: eg, surgery resulting in complicated lens placement (such as anterior chamber intraocular lens implant (IOL); phakie IOL; sulcus IOL; aphakia, etc) or intraoperative complications (eg such as a posterior capsular tear [with or without vitreous loss], substantial iris trauma, etc) Note: history of uncomplicated cataract surgery is not an exclusion. Updated the statistical analyses as follows: Intraocular pressure change from baseline will be analyzed using a mixed-effects model repeated

## Section Revision Rationale measures (MMRM) approach. The model will include the fixed effects of treatment; IOP time-matched change from baseline IOP stratification; visit ( as the response variable and treatment, timepoint (Hours 0 and 2 at each visit of Weeks 2, 6, and 12),; hour; the two way interaction between treatment and each of hour and visit; and the three way treatment-bytimepoint interaction between treatment, hour, and visit and baseline IOP stratification as fixed effects. Unstructured covariance matrix will be used for repeated measures on the same patient; if the model with unstructured covariance matrix fails to converge, multiple imputation (MI) will be implemented before MMRM. For the United States Food and Drug Administration (US FDA), the primary efficacy variable will be the study eye time matched IOP. The primary analysis will be based on Weeks 2, 6, and 12 using the ITT population. Specifically, the following analysis will be performed: time matched IOP will be analyzed using an MMRM approach based on the same model as described for the primary efficacy analysis of timematched IOP change from baseline. Sample Size Calculation: The sample size calculation is based on the primary efficacy analysis of the time matched IOP for US FDA review because the sample size based on the primary efficacy analysis for other regions is expected to be smaller. Table 2



| Section | Revision | Rationale |
|---|---|---|
| | target) tissues with concentrations in the bulbar conjunctiva, eyelid margin, and periorbital fat significantly higher than those observed in the iris-ciliary body. In contrast, following administration of a single. Bimatoprost SR implant at 15 µg, bimatoprost and bimatoprost acid concentrations were either below the limit of quantitation (BLQ) or near the detection limit in bulbar conjunctiva, eyelid margin, and periorbital fat while the highest bimatoprost and bimatoprost acid concentrations were observed in the target tissue, the iris ciliary body. Retinal concentrations were BLQ following both topical and Bimatoprost SR administration. | |
| Section<br>1.3.3 | Study 192024-041D is an ongoing was a Phase 1/2, pairedeye comparison evaluating the safety and efficacy of 4 dose strengths of Bimatoprost SR (6 µg, 10 µg, 15 µg, or 20 µg [2 × 10 µg implants]), as single or repeat administration in one eye (study eye), versus the use of topical LUMIGAN® 0.03% in the fellow eye (nonstudy eye). The objective of this study is was to evaluate the safety and IOP-lowering efficacy of Bimatoprost SR in patients with OAG. | Updated information from recently completed study |
| | As of March 2015, a total of 109 patients had received a single administration; and as of June 2015, 24 patients had received a repeat administration of Bimatoprost SR. Based on a review of the efficacy data as of March 2015, a A trend in dose response has been was observed across the 4 dose strengths that were tested. Available d Data suggest that the implant may provide topical prostaglandin analog-like efficacy up to 3 to 4 months post-implantation in the majority of patients. Data following the second administration in the redosed patients showed similar IOP lowering to that observed following the first administration of Bimatoprost SR. | |
| | As of March 2015, Bimatoprost SR has shown showed an acceptable safety profile with single and repeat administrations in ongoing s Study 192024-041D. Most adverse events were ocular, mild or moderate in severity, occurred within the first \$ 2 days after Bimatoprost SR administration, and were considered related to the study drug administration procedure. There has shown were no reports of serious study drug-related adverse events, and no new safety concerns has shown were observed after the second treatment. Please refer to the Investigator's Brochure for details on reported safety findings. | |
| Section 3 | The study will be conducted at approximately 1650 sites globally. | Revised to reflect actual number of sites |
| Section<br>4.1 | Enrollment of approximately 600 patients in total at approximately 150 160 sites, with approximately 200 patients per group, is planned to ensure 180 completed patients per group, assuming a premature discontinuation rate of 10%. | Revised to reflect actual number of sites |
| Section<br>4.2 | The study population consists of patients with OAG or OHT and an open iridocorneal angle inferiorly by clinical | Revised for consistency with updated inclusion criteria |

#### Section Revision Rationale gonioscopy in the study eye, and OAG or OHT in the fellow eye, where both eyes require IOP-lowering medication. The eye that meets the entry criteria (Sections 4.3 and 4.4) will be selected as the study eye. If both eyes meet the entry criteria (including iridocorneal angles that have been confirmed as qualified by the Reading Center anterior segment optical coherence tomography [AS-OCT assessment]), the eye with the higher IOP at Baseline Hour 0 will be selected as the study eye. If both eyes have the same IOP, then the right eye will be designated as the study eye. Angle qualification will be independently confirmed as being qualified by 2 ophthalmologists, and endothelial cell density qualification for study entry will be determined by the Reading Center based on AS OCT and specular microscopy assessment respectively (see Protocol Procedure Manual for details). Patients With Sickle Cell Trait or Disease Section 4.2.1 Based on the ongoing safety 4.2.1 monitoring of the 192024-091 and At screening all patients will be tested for sickle cell trait or 192024-092 studies, no increased disease. Patients with sickle cell trait or disease (or other risk of hyphema or microhyphema hemoglobinopathies) may be enrolled at the discretion of with sickle cell traits or sickle cell the investigator based on an individual risk-benefit disease is confirmed. There are assessment. Because of a slightly higher risk of IOP 400+ patients had at least one elevation and intraocular complications in the setting of a Bimatoprost SR injection in the microhyphema, patients with these disorders must may 2 studies (estimated based on 1:1:1 undergo optional additional safety monitoring ratio), there is only one report of (biomicroscopy and IOP measurements) after microhyphema in a NON-sickle cell injection/Sham injection at the investigator's discretion (as patient. No anterior chamber safety outlined in see Section 8.4). Additional information about concerns reported in the 14 sickle the Bimatoprost SR experience in patients with sickle trait cell or traits patients. is provided in the Investigator's Brochure. Section 43



| Section | Revision | Rationale |
|---|---|---|
| Section<br>5.7 | Investigational medicinal product must be stored as described in the Investigator's Brochure Investigational medicinal product must be stored at a room temperature representing a usual and customary working environment, as described in the Protocol Procedure Manual. | With the product being under<br>development, the current details on<br>the storage conditions will be<br>reflected in the Investigator's<br>Brochure. |
| Section 5.9.4 | Note: Patients with sickle cell disease or trait (or other hemoglobinopathies) will be expected to may undergo optional biomicroscopy and IOP examination in both eyes 4 hours after each Bimatoprost SR administration (or Sham administration). This optional IOP examination is for postoperative purposes only, and as such does not require a masked, 2-person reading method. The IOP should be taken only once to avoid excessive postadministration (or Sham administration) manipulation of the eye, and should be taken by the investigator (or other unmasked, qualified personnel). This postadministration (or Sham administration) examination may be performed using a Goldmann applanation tonometer or a hand-held tonometer. (See the Study Procedure Manual for details.) | Based on the ongoing safety monitoring of the 192024-091 and 192024-092 studies, no increased risk of hyphema or microhyphema with sickle cell traits or sickle cell disease is confirmed. There are 400+ patients had at least one Bimatoprost SR injection in the 2 studies (estimated based on 1:1:1 ratio), there is only one report of microhyphema in a NON-sickle cell patient. No anterior chamber safety concerns reported in the 14 sickle cell or traits patients. |
| Section<br>6.2 | Hematology, blood chemistry, and urinalysis: Blood and urine samples will be collected for blood chemistry and hematology panels (including sickle cell testing by local laboratories) and urinalysis. | Based on the ongoing safety monitoring of the 192024-091 and 192024-092 studies, no increased risk of hyphema or microhyphema with sickle cell traits or sickle cell disease is confirmed. There are 400+ patients had at least one Bimatoprost SR injection in the 2 studies (estimated based on 1:1:1 ratio), there is only one report of microhyphema in a NON-sickle cell patient. No anterior chamber safety concerns reported in the 14 sickle cell or traits patients. |



| Section | Revision | Rationale |
|---|---|---|
| | been unmasked after each lock will no longer be involved directly in any ongoing masked study conduct. Another statistician, who is still masked to study treatment, will assume these responsibilities until the next lock. Unmasked data handling and appropriate data and results access will be specified prior to each lock. | |
| Section<br>7.2 | To avoid confounding of efficacy data, IOP measurements obtained after initiating the use of nonstudy IOP-lowering medication in an eye will be treated as missing for that eye excluded from the calculation of the summary statistics and the statistical analyses for that eye but raw values will be presented in the listings. | Updated text for clarity. |
| Section<br>7.3.1 | Intraocular pressure change from baseline will be analyzed using a mixed-effects model repeated measures (MMRM) approach. The model will include the fixed effects of treatment; IOP time-matched change from baseline IOP stratification; visit (as the response variable and treatment, timepoint (Hours 0 and 2 at each visit of Weeks 2, 6, and 12); hour; the two way, treatment-by-timepoint interaction, between treatment and each of hour and visit; and the three-way interaction between treatment, hour, and visit baseline IOP stratification as fixed effects. Unstructured covariance matrix will be used for repeated measures on the same patient; if the model with unstructured covariance matrix fails to converge, multiple imputation (MI) will be implemented before MMRM. The details of the model specifications will be provided in the analysis plan. | Updated text for clarity. |
| Section<br>7.3.2 | Secondary efficacy analyses comparing each Bimatoprost SR dose strength and timolol to test the no-difference null hypothesis will be performed at scheduled visits (Weeks 2, 6, and 12) and hours for (1) time matched IOP and (2) timematched IOP change from baseline. The analysis of time matched IOP will be similarly performed as described above with time matched IOP replacing time-matched IOP change from baseline in the analysis model. | Updated text for clarity. |
| Section<br>7.6 | For the US FDA review, the primary efficacy variable will be the study eye time matched IOP. | Updated text for clarity. |
| | For each Bimatoprost SR dose strength which demonstrates efficacy (clinical noninferiority) as described in the primary efficacy analyses, secondary efficacy analyses comparing the Bimatoprost SR dose strength and timolol to test the no-difference null hypothesis will be performed at scheduled visits (Weeks 2, 6, and 12) and hours for time matched IOP. | |





# **ALLERGAN**

### Protocol 192024-091 Amendment 2

Date (DD/MMM/YYYY)/Time (PT) Signed by: Justification